Statistical Analysis Plan J2G-OX-JZJE Final Version

A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of LOXO-292

NCT05469100

Approval Date: 03-Jun-2019



- **16.1.9 Documentation of Statistical Methods**
- 16.1.9.1 Statistical Analysis Plan

# Statistical Analysis Plan

A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of LOXO-292

Protocol No: LOXO-RET-18023 Final Protocol Date: 22 October 2018 Amendment 1 Date: 04 December 2018 Amendment 2 Date: 09 January 2019 Amendment 3 Date: 09 May 2019 Compound Name: LOXO-292

> Celerion Project CA25886 Final Version 1.0 Date: 23 May 2019

Loxo Oncology, Inc. 701 Gateway Boulevard, Suite 420 South San Francisco, California 94080, USA

Celerion 100 Alexis-Nihon Boulevard, Suite 360, Montreal, QC H4M 2N8, Canada

# Statistical Analysis Plan Signature Page

Compound Name: LOXO-292

Protocol: LOXO-RET-18023

Study Title: A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Evaluate the

Effect of Renal Impairment on the Pharmacokinetics of LOXO-292

Issue Date: 23 May 2019



# **Table of Contents**

| 1.2 | INTE | RODUCTION | 52 |
|---|---|---|---|
| 2.2 | OBJI | ECTIVES AND ENDPOINTS | 52 |
| | 2.12 | Objectives | 52 |
| | | Endpoints | |
| 3.? | STU | DY DESIGN | 62 |
| 4.? | ANA | LYSIS POPULATIONS | 82 |
| | 4.12 | Analysis Populations | 82 |
| | 4.22 | Preliminary Data and Interim Analysis | 82 |
| 5.2 | TRE | ATMENT DESCRIPTIONS | 82 |
| 6.2 | PHA | RMACOKINETIC ANALYSIS | 9? |
| | 6.12 | Measurements and Collection Schedule | 92 |
| | 6.22 | Bioanalytical Method | 102 |
| | 6.32 | Investigational Product and PK Analyte Information of LOXO-292 | |
| | | Pharmacokinetic Concentrations. | 102 |
| | 6.52 | Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292 | 11 |
| | | 6.5.12 Plasma Pharmacokinetic Parameters | |
| | | 6.5.22 Unbound Plasma LOXO-292 Pharmacokinetic Parameters | 122 |
| | | 6.5.32 Urine Pharmacokinetic Parameters | 142 |
| | 6.62 | Data Summarization and Presentation | 152 |
| | 6.72 | Statistical Analysis of PK Parameters | 172 |
| | | 6.7.12 Primary Analysis | 172 |
| | | 6.7.22 Analysis of Covariance | 182 |
| | | 6.7.32 Additional Analysis | 192 |
| 7.2 | SAF | ETY | 192 |
| | | Subject Discontinuation | |
| | 7.22 | Demographics | 202 |
| | 7.32 | Adverse Events. | 202 |
| | 7.42 | Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis) | 22 |
| | 7.52 | Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and | |
| | 7.62 | Temperature) | |
| | 7.00 | correction]) | 232 |
| | 7.72 | Concomitant Medications | |
| | 7.82 | Physical Examination. | 242 |
| <b>Ω</b> ΓΙ | STIM | IMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 245 |

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886

| 9.2 | SUMMARY TABLES AND FIGURES | 24 |
|-----|--------------------------------------------|----|
| | 9.12 In-text Summary Tables and Figures | 24 |
| | 9.22 Section 14 Summary Tables and Figures | |
| | 9.32 Section 16 Data Listings | |
| 10. | TABLE AND FIGURE SHELLS | 42 |
| | 10.12 In-text Table Shells | 43 |
| | 10.22 Figures Shells | 50 |
| | 10.32 Post-text Table Shells | |
| 11. | LISTING SHELLS | 89 |

## 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from study LOXO-RET-18023. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within the protocol or after the locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by Loxo Oncology, Inc., will be considered out of scope and will be described in the CSR as needed.

#### 2. OBJECTIVES AND ENDPOINTS

## 2.1 Objectives

## **Primary:**

To compare the plasma pharmacokinetics (PK) of LOXO-292 following administration in subjects with varying degrees of renal impairment (RI) (i.e., mild, moderate, and severe) compared to healthy matched control subjects.

#### **Secondary:**

- 1. To evaluate the safety and tolerability of LOXO-292 in subjects with RI.
- 2. To compare the urine PK of LOXO-292 following administration in subjects with varying degrees of RI (i.e., mild, moderate, and severe) compared to healthy matched control subjects.

# 2.2 Endpoints

## **Pharmacokinetics:**

The following PK parameters will be calculated for LOXO-292 in plasma, as appropriate: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, t½, CL/F, and Vz/F.

The following PK parameters will be calculated for unbound LOXO-292: AUC0-t,u, AUC0-inf,u, Cmax,u, CL/F,u, and Vz/F,u.

The following PK parameters will be calculated for LOXO-292 in urine, as appropriate, in all cohorts: Ae, Fe, and CLr.

## Safety:

Safety endpoints will include 12-lead electrocardiograms (ECGs), physical examinations, vital signs, clinical laboratory tests, and adverse events (AEs).

## 3. STUDY DESIGN

This is a non-randomized, open-label, parallel-cohort, multiple-site, single-dose study to compare the PK of LOXO-292 in subjects with mild, moderate, and severe RI compared to healthy matched control subjects matched 1:1 for age, body mass index (BMI), and sex.

Up to 48, adult male and female subjects will be enrolled.

# **Subjects with RI:**

Up to 24 subjects with RI will be enrolled as follows:

Up to eight (8) subjects with mild RI.

Up to eight (8) subjects with moderate RI.

Up to eight (8) subjects with severe RI.

# **Healthy Matched Control Subjects:**

Up to 24 healthy subjects will be enrolled to ensure that each subject in the RI cohorts will be matched with a healthy subject based on sex, age ( $\pm$  10 years), and BMI ( $\pm$  20%). An individual healthy subject may be matched to one subject from each of the RI cohorts (mild, moderate, and severe) providing matching criterion are met, and such that each healthy subject may be matched to a maximum of 3 subjects with RI. However, no healthy subject can be matched to more than one subject in any single RI cohort.

Screening of subjects will occur within 28 days prior to LOXO-292 dosing.

On Day 1, subjects will receive a single oral dose of LOXO-292. Plasma and urine samples will be collected predose (if possible) and through 168 hours postdose for healthy subjects and subjects with RI for LOXO-292 PK assessment.

Assignment to a renal function panel will be as follows:

| Cohort | Renal Function | eGFR (mL/min/1.73m <sup>2</sup> ) * |
|--------|-------------------------|-------------------------------------|
| 1 | Healthy Matched Control | ≥ 90 ** |
| 2 | Mild | 60 ≤ eGFR < 90 |

| Cohort | Renal Function | eGFR (mL/min/1.73m²) * |
|---|---|---|
| 3 | Moderate | 30 ≤ eGFR < 60 |
| 4 | Severe (not on dialysis) | < 30 |
| | subjects with RI and healthy-n the mean of the eGFR obtained historical values within a 3-mo historical measurement is avait sample will be taken during the apart) and the mean of the two Baseline eGFR for cohort assis recorded for each measurement baseline value must fall within each cohort (i.e., healthy, mild categorize subjects' renal impa ** For healthy-matched control actual creatinine clearance con collection may be used in place | Disease (MDRD) equation at 1 be obtained for all subjects (i.e., natched control subjects) by taking d from Screening and from onth period from Screening. If no lable, a second Screening eGFR e Screening period (≥ 14 days values will be used as the gnment. Individual eGFR values at contributing to the subject mean a the specified eGFR ranges for 1, moderate, and severe) to airment status. |

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

Subjects may be replaced at the discretion of the Sponsor.

Subjects will be housed in the clinical research unit (CRU) from Check-in (Day -1), at the time indicated by the CRU, until after completion of the Day 8 (End of Treatment [EOT]) or Early Termination (ET) study procedures. EOT is defined as the day on which the subject is released from the CRU, following all study procedures.

The CRUs will contact all subjects who received LOXO-292 (including subjects who terminate from the study early) at the End of Study (EOS,) by a follow up phone call (FU). The EOS/FU phone call will be performed 7 days ( $\pm$  2 days) after the EOT visit or ET visit to determine if any study drug-related adverse event (AE) or serious adverse event (SAE) has occurred since the EOT or ET visit.

## 4. ANALYSIS POPULATIONS

# 4.1 Analysis Populations

## **Safety Population**

All subjects who received a dose of the study drug will be included in the safety evaluations.

# Pharmacokinetic Population

Samples from all subjects will be assayed even if the subjects do not complete the study. All subjects who comply sufficiently with the protocol and display an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses.

Data for each subject will be included in the summary statistics and statistical comparisons of PK parameters with the exceptions described as follows:

- Data from subjects who experience emesis at or before 2 times median Tmax for LOXO-292 during the PK sampling period of the study may be excluded from the summary statistics and from the statistical comparison of PK parameters.
- All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when subjects are assigned to analysis populations.

Any subject or data excluded from the analysis will be identified, along with their reason for exclusion, in the CSR.

# 4.2 Preliminary Data and Interim Analysis

No formal interim analysis is planned.

#### 5. TREATMENT DESCRIPTIONS

LOXO-292 will be supplied as 80 mg capsules.

Subjects will receive a single oral dose of 160 mg LOXO-292 (2 x 80 mg capsules) on Day 1 following a fast from food of at least 2 hours (not including water), with approximately 240 mL of water, followed by a fast from food (not including water) for at least 1 hour postdose.

Subjects will be instructed not to crush, split, or chew LOXO-292.

**Table 5.1 Cohort Description** 

| Cohort | Short Description (text, tables<br>headers, footers, figures,<br>listings, SAS output) | Description |
|---|---|---|
| Mild | Subjects with Mild RI (n = 8) | Administration of a single oral dose of 160 mg LOXO-292 to subjects with mild renal impairment following a 2-hour fast. |
| Moderate | Subjects with Moderate RI (n = 8) | Administration of a single oral dose of 160 mg LOXO-292 to subjects with moderate renal impairment following a 2-hour fast. |
| Severe | Subjects with Severe RI (n = 8) | Administration of a single oral dose of 160 mg LOXO-292 to subjects with severe renal impairment following a 2-hour fast. |
| Healthy | Healthy Matched Control<br>Subjects<br>(n = 8 up to 24) | Administration of a single oral dose of 160 mg LOXO-292 to healthy match control subjects following a 2-hour fast. |

# 6. PHARMACOKINETIC ANALYSIS

# 6.1 Measurements and Collection Schedule

# Plasma

Blood samples for PK assessment of LOXO-292 will be taken at the following time points:

CCI

#### Urine

Urine will be collected at predose (spot collection) and during the following postdose intervals:

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there are any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. The exclusion of data will be made in agreement between the Sponsor and Celerion. All deviations and excluded data will be provided and discussed in the CSR.

# 6.2 Bioanalytical Method

Plasma and urine concentrations of LOXO-292 will be determined using a liquid chromatography-tandem mass spectrometry (LC-MS/MS) method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Alturas Analytics, Inc. (Moscow, Idaho, USA). The analytical rang CCI

Samples that contain concentrations greater than 1000 ng/mL may be diluted up to CCI, if necessary, to be within the quantification range. The analytical range CCI Samples of urine that contain concentrations greater than CCI may be diluted, if necessary, to be within the quantification range.

# 6.3 Investigational Product and PK Analyte Information of LOXO-292

LOXO-292 has a molecular weight of approximately CC . LOXO-292 will be supplied as a simple blend with excipients containing 80 mg of drug substance (freebase) in a hard gelatin capsule.

# 6.4 Pharmacokinetic Concentrations

Plasma and urine concentrations of LOXO-292 as determined at the collection times and per the bioanalytical method described in Sections 6.1 and 6.2, respectively, will be used for the calculation of the plasma LOXO-292 PK parameters.

# 6.5 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292

# 6.5.1 Plasma Pharmacokinetic Parameters

The appropriate noncompartmental PK parameters will be calculated from the total plasma LOXO-292 concentration-time data using Phoenix® WinNonlin® Version 7.0 or higher. Actual sample collection times, relative to the administration time of LOXO-292, will be used in the calculations of the PK parameters. All total plasma PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Total Plasma Pharmacokinetic Parameters to be Calculated for LOXO-292

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t | Area under the concentration-time curve for LOXO-292 concentration from time 0 to the time of the last observed non-zero concentration | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| AUC0-inf | Area under the concentration-time curve for LOXO-292 concentration from time 0 extrapolated to infinity | Calculated as AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration |
| AUC%extrap | Percent of AUC0-inf extrapolated | Calculated as<br>(1 -<br>AUC0-t/AUC0-inf)*100 |
| Cmax | Maximum observed LOXO-292 concentration | Taken directly from bioanalytical data |
| Tmax | The time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |
| Kel | Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time | Calculated as the negative of the slope of a linear regression of the log(concentration)-time for all concentrations >LLOQ during the terminal elimination phase |
| t½ | Apparent first-order terminal elimination half-life | Calculated as 0.693/Kel |

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| CL/F | Apparent total plasma clearance after oral (extravascular) administration | Calculated as<br>Dose/(AUC0-inf) |
| Vz/F | Apparent volume of distribution of LOXO-292 during the terminal elimination phase after extravascular administration | Calculated as Dose/(AUC0-inf x Kel) |

Pharmacokinetic parameters will not be calculated for subjects with fewer than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the statistical analysis.

For the calculation of the PK parameters, plasma concentrations below the limit of quantitation (BLQ) prior to the first quantifiable concentration will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

The Kel will be determined using linear regressions composed of least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of t½, AUC0-inf, AUC%extrap, CL/F, Vz/F are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated parameters (t½, AUC0-inf, AUC%extrap, CL/F, and Vz/F) may not be presented as judged appropriate and in accordance with Celerion SOPs.

## 6.5.2 Unbound Plasma LOXO-292 Pharmacokinetic Parameters

An analysis to determine the unbound plasma LOXO-292 PK parameters will be conducted. The fraction of unbound (fu) LOXO-292 in plasma for each subject will be estimated via an ex vivo protein binding analysis using a predose plasma sample. Unbound plasma concentrations of LOXO-292 will be calculated by multiplying the measured plasma concentrations by the fraction unbound of each subject (Cu = measured concentration x fu) at each sampling time point for that subject. The following unbound PK parameters using the individual Cu values and actual sampling times using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 7.0 or higher:

Table 6.2. Noncompartmental Plasma Pharmacokinetic Parameters to be Calculated for Unbound LOXO-292

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t,u | Area under the concentration-time curve for unbound LOXO-292 concentration from time 0 to the time of the last observed non-zero | Calculated using the<br>Linear Trapezoidal with<br>Linear Interpolation<br>Method |
| AUC0-inf,u | Area under the concentration-time curve for unbound LOXO-292 concentration from time 0 extrapolated to infinity | Calculated as AUC0-t,u + (Clast,u/Kel,u) where Clast is the last observed/measured unbound concentration |
| Cmax,u | Maximum observed unbound LOXO-292 concentration | Taken directly from<br>unbound plasma<br>concentration of<br>LOXO-292 |
| Kel,u | Apparent terminal elimination rate constant; represents the fraction of unbound drug eliminated per unit time | Calculated as the negative of the slope of a linear regression of the log(unbound concentration)-time for all unbound concentrations >LLOQ during the terminal elimination phase |
| CL/F,u | Apparent total plasma clearance of unbound LOXO-292 after extravascular (oral) administration | Calculated as Dose/(AUC0-inf,u) |
| Vz/F,u | Apparent volume of distribution of unbound LOXO-292 during the terminal elimination phase after extravascular administration | Calculated as Dose/(AUC0-inf,u x Kel,u*) |

<sup>\*</sup> The same timepoints selected for the calculation of Kel will be selected for the calculation of Kel,u. Kel,u will be calculated in WinNonLin but will not be presented in tables.

Unbound PK parameters will not be calculated for subjects with fewer than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the statistical analysis.

For the calculation of the unbound PK parameters, plasma concentrations BLQ prior to the first quantifiable concentration will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

The Kel,u will be determined using linear regressions composed of least 3 data points. The Kel,u will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax,u is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel,u interval is not assigned, the values of t½,u, AUC0-inf,u, CL/F,u, and Vd/F,u are considered not calculable and will not be reported. Wherever the resulting t½,u is more than half as long as the sampling interval, the Kel,u values and associated parameters (t½,u, AUC0-inf,u, CL/F,u, and Vd/F,u) may not be presented as judged appropriate and in accordance with Celerion SOPs.

#### 6.5.3 Urine Pharmacokinetic Parameters

The following PK parameters will be calculated from urine LOXO-292 data using SAS® Version 9.3 or higher. All urine PK parameters included in the protocol are listed in Table 6.3 below, and are defined as appropriate for study design.

Table 6.3. Noncompartmental Urine Pharmacokinetic Parameters to be Calculated for LOXO-292

| Label to be<br>Used in Text,<br>Tables and<br>Figures | Definition | Method of Determination |
|---|---|---|
| Aet1-t2 | Amount of unchanged LOXO-292 excreted during urine collection interval from t1 to t2; the collection | Calculated as: Urine LOXO-292 concentration * urine volume Note: If the amount of urine excreted was captured in the CRF as urine weight (g), it will be converted to volume (mL) using the assumed density of 1 g/mL. |

| Label to be<br>Used in Text,<br>Tables and | | |
|---|---|---|
| Figures | Definition | Method of Determination |
| Ae0-t | Total amount of LOXO-292 excreted unchanged in the urine over the entire urine collection period (0-t hours) | Calculated as: The sum of the individual Aet1-t2 (urine LOXO-292 concentration * urine volume) over the entire urine collection interval Note: If the amount of urine excreted was captured in the CRF as urine weight (g), it will be converted to volume (mL) using the assumed density |
| CLr | Renal clearance | of 1 g/mL. Calculated as: Ae(t1-t2)/AUC(t1-t2) Where t1-t2 is the longest interval of time during which Ae and AUC are both obtained. |
| Fe | The percent of dose excreted unchanged into urine from time 0 to the time at the end of the urine collection interval | Calculated as: 100*[Ae0-t]/Dose Where Ae0-t is the cumulative amount of LOXO-292 excreted unchanged in the urine over the entire urine collection period (0-t hours) and dose is the dose of the free base LOXO-292 |

For the calculation of the urine PK parameters, urine data BLQ concentrations will be treated as 0. See Section 6.6 for further information on missing urine data.

# 6.6 Data Summarization and Presentation

All LOXO-292 PK concentrations and PK parameters descriptive statistics will be generated using SAS® Version 9.3 or higher.

The total and unbound plasma concentrations of LOXO-292 will be listed and summarized by cohort and time point for all subjects in the PK Population. For the protein binding assay, the buffer chamber (BC) and plasma chamber (PC)

concentrations, % recovery, and fraction unbound will be listed and summarized by cohort for all subjects in the PK Population. The urine concentrations of LOXO-292 will be listed and summarized by cohort and collection-intervals for all subjects in the PK Population.

Plasma and urine concentrations of LOXO-292 will be presented with the same level of precision as received from the bioanalytical laboratory. Unbound plasma concentrations of LOXO-292 will be presented with the same level of precision as received from the bioanalytical laboratory. Data from the protein binding assay will be presented with the same level of precision as received from the bioanalytical laboratory.

Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points and collection intervals. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual total and unbound plasma concentration-time profiles will be presented on linear and semi-log scales. Linear mean plots will be presented with and without SD. Urine data will be graphically summarized with mean and individual cumulative amounts of LOXO-292 excreted (Ae0-t) and cumulative % dose excreted unchanged versus end of collection interval, on linear plots (with and without SD for mean).

Total and unbound plasma LOXO-292 PK parameters will be listed and summarized by cohort for all subjects in the PK Population. PK parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax and t½, which will be presented with 2 decimal places. Summary statistics (n, Mean, SD, CV%, SEM, minimum, median, maximum, geometric mean [Geom Mean], geometric CV% [Geom CV%], and 95% CI Geom Mean [presented for AUC0-t, AUC0-inf and Cmax only]) will be calculated for total and unbound plasma LOXO-292 PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

For urine data, in cases where a subject was unable to void during a given interval, the urine volume for that interval will be set to zero, labeled as "UTV" (i.e., "unable to void"), and footnoted accordingly. All urinary parameters requiring volume in their calculation, for that interval only, will be set to zero. The cumulative amount excreted for that interval will be calculated as the previous cumulative amount plus 0. If a sample was collected, but volume was not recorded or only a partial volume was recorded, the urine volume for this that interval will be set to missing and footnoted accordingly. All urinary parameters requiring volume in their calculation, for that interval only, will be set to missing. The cumulative amount excreted for that interval

and all intervals thereafter, including the total cumulative amount excreted, are not calculable and will be set to missing. With the exception of those parameters set to missing, no parameters will be excluded from summary statistics. Furthermore, only results up to the missing interval will be included in summary statistics and in presentation of cumulative urinary excretion plots. Urine concentration results from and beyond the missing interval will be listed in the table and summarized accordingly.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and parameter output,
- mean/median/Geom Mean in one more level of precision than minimum/maximum,
- SD/SEM in one more level of precision than mean/median/Geom Mean,
- n will be presented as an integer, and
- CV%/ Geom CV% will be presented to the nearest tenth.
- 95% CI Geom Mean will be presented with 2 decimals.

# 6.7 Statistical Analysis of PK Parameters

# 6.7.1 Primary Analysis

A comparison of natural-log (ln)-transformed PK parameters (total: AUC0-t, AUC0-inf, and Cmax, and unbound: AUC0-t,u, AUC0-inf,u, and Cmax,u) will be made to evaluate the effect of renal function group on the PK of a single dose of LOXO-292. Since the comparison groups of subjects are independent in terms of degrees of RI and dependent based on the matching criteria, paired t-tests will be performed, using PROC TTEST of SAS®, to assess the differences in PK parameter between each hepatic impairment group versus the corresponding healthy matched control group with respect to 1 to 1 matching. Geometric mean ratios (GMRs) and ninety percent (90%) confidence intervals (CIs) for the ratios will be derived by exponentiation of the mean difference and the CIs obtained for the difference in mean between each renal function cohort and the matching healthy control group.

The paired t-test analysis for each PK parameter will be performed using the following SAS® code for each renal function cohort and its corresponding healthy matched control group:



# CCI

RUN;

Programmer note: The paired t-test will be performed for each renal function group and the subset of corresponding healthy matched control subjects separately. LPKri refers to the set of ln-transformed PK parameters for the subjects in the renal impaired function group of interest (i.e., Mild, Moderate, or Severe) and LPKhealthy refers to the ln-transformed PK parameters for the set of corresponding matching healthy control subjects.

# 6.7.2 Analysis of Covariance

An analysis of covariance (ANCOVA) will also be performed on the In-transformed PK parameters (total: AUC0-t, AUC0-inf, and Cmax, and unbound: AUC0-t,u, AUC0-inf,u, and Cmax,u) of LOXO-292 to evaluate the effect of various degrees of RI on the PK of LOXO-292. The ANCOVA model will contain a categorical factor of population for subjects with various degrees of RI (mild, moderate, severe, and healthy matched control subjects), a categorical covariate (sex), and continuous covariates (age and BMI).

Ratios of least-squares means (LSMs) and 90% CIs of ratios will be calculated using the exponentiation of the difference between two cohort LSMs and the corresponding CIs from the ANCOVA analyses on the ln-transformed AUC0-t, AUC0-inf, and Cmax and the corresponding unbound parameters, AUC0-t,u, AUC0-inf,u, and Cmax,u. These ratios will be expressed as a percentage relative to the healthy matched control cohort. Geometric LSM, GMRs, and 90% CIs will be presented.

The ANCOVA analysis will be performed using the following SAS® code:



Programmer Note: The coefficients in the estimate statements presented above assume that the following decodes will be used for cohort in the database: Mild RI = A, Moderate RI = B, Severe RI = C, Healthy Matched Control = D. Please confirm these coefficients with the Biostatistician prior to data analysis.

# 6.7.3 Additional Analysis

The relationship between LOXO-292 PK parameters (i.e., Cmax and AUC, total and unbound) and measures of renal function (such as eGFR and CLcr) will be examined in an exploratory manner via a graphically linear regression approach. The PK parameters will be the dependent variable and show on y-axis and measurements for renal impairment will be independent variables and show on the x-axis. The regression equation with slope and intercept, the r-square, and the p-value for slope will be presented in the graphs as footnotes.

If data permits and judged necessary, an exploratory analysis will be performed to assess the relationship between LOXO-292 PK and renal impairment and the effect of covariates (age, BMI, and gender) using an appropriate approach.

#### 7. SAFETY

No inferential statistics are to be performed for the safety analysis.

All clinical safety and tolerability data will be listed by cohort, subject and assessment time points, chronologically. This will include unscheduled assessments (including rechecks) and ET records.

Continuous variables will be summarized using n, mean, SD, minimum, median, and maximum. Frequency counts will be reported for categorical data when appropriate. The level of precision will be presented as follows: "n" as an integer, minimum/maximum in same precision as in the database, mean/median in one more precision level than minimum/maximum, and SD in one more precision level than mean/median. Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

When change from baseline is calculated, baseline is the last scheduled or unscheduled assessment before dosing on Day 1, whichever is later. Unscheduled assessments and ET measurements taken after dosing will not be used in the summarization.

Note: The term 'unscheduled' assessment used in this SAP may also refer to recheck assessments.

# 7.1 Subject Discontinuation

Subjects will be summarized by the number of subjects enrolled, completed, and discontinued from the study with discontinuation reasons by cohort and overall. Discontinuation data will be listed by-subject.

# 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) by cohort and over all the study. Weight, height and body mass index are summarized at screening. Age will be derived from the date of birth to the date of dosing. Frequency counts will be provided for categorical variables (race, ethnicity, and sex) by cohort and over all the study. A by-subject listing will also be provided.

# **7.3** Adverse Events

All AEs occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 21.1.

Each AE will be graded, by the clinical site, on the National Institution of Health's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) 5-point severity scale (Grade 1, 2, 3, 4 and 5). Not all grades are appropriate for all AEs. Therefore, some AEs are listed within the CTCAE with fewer than 5 options for grade selection.

The following clinical descriptions of severity for each AE are based on the following general guideline [CTCAE Nov2017]:

**Table 7.3: Adverse Event Severity Level and Description** 

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |

| Grade | Description |
|---------|----------------------|
| Grade 5 | Death related to AE. |

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

Similarly, the causal relationship of the study drug to the AE will be described as Related or Not related to study drug (LOXO-292). All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, cohort, severity grade, relationship to study drug, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an undesirable event not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. Each TEAE will be attributed to the treatment based on Investigator (or designee) judgment as well as on its onset date and time. If an AE has a change in severity grade, the original AE will be given a resolution date and time of the time of severity grade increase or decrease and a new AE record will be initiated with the new severity grade, and the new AE record will use the resolved date/time of the previous record as the onset date/time. If the severity grade of an AE remains the same, the AE will be kept open through to resolution.

If the onset date and/or time of an AE is/are missing, the AE will be treated as a TEAE, unless the onset date of the AE is known to have occurred prior to dosing. TEAEs will be tabulated by system organ class and preferred term. Summary tables will include the number of subjects reporting the AE and as a percent of the number of subjects dosed by cohort and overall. In addition, the number of AEs will be summarized. For an AE with multiple changes in severity, a new record with severity less or equal to its maximum severity will not be included in the adverse event summary tables. Tables will also be presented by severity grade and relationship to study drug. If a subject experienced the same TEAE at more than once with different level of severity grade, only the most severe one will be counted. Similarly, if a subject experienced the same TEAE more than once with different level of drug relationship, only the one most closely related to the study drug will be counted.

Should any serious adverse events (SAEs) occur during the study, the SAEs will be displayed in a table and a narrative included in the Clinical Study Report.

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications and not bedridden.□

# 7.4 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis)

All clinical laboratory test results will be presented in by-subject data listings, however, only serum chemistry, hematology, coagulation and urinalysis values will be summarized. Given that this study was conducted at multiple sites, by-subject data listings will be provided in conventional units and international system of units (SI units). Summary tables will be provided in SI units.

Hematology, coagulation, serum chemistry and urinalysis tests will be conducted at the following time points:

**Table 7.4 Lab Test Time Points** 

| Day |
|------------------------------------------|
| Screening* |
| Day -1* |
| Day 2 |
| Day 5 |
| Day 8** |
| * performed following a fast of at least |
| 12 hours |
| ** performed at EOT or prior to ET |

Out-of-normal range flags will be presented in the clinical laboratory listings as recorded in the database. The reference ranges used during the study will be provided in conventional and SI units by study site in Appendix 16.1.10.1. Out-of-range values and unscheduled results will be listed. Results that are indicated as CS by the PI (either in the PI flag or in PI comments) will be listed in the table.

For all laboratory values that are numeric, descriptive statistics (n, mean, SD, minimum, median, and maximum) will be presented for each laboratory test by cohort and time point. Change from baseline will also be summarized. Postdose unscheduled assessments and ET results will not be summarized.

For each laboratory test, a shift table will be developed comparing the frequency of the results at baseline (above normal, normal, or below normal) to postdose results. For urinalysis tests, the categories are normal and outside normal.

Baseline is the last non-missing predose measurement prior to dosing (Day -1), including unscheduled assessments.

# 7.5 Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and Temperature)

Vital signs will be performed at the following time points:

**Table 7.5 Vital Signs Time Points** 

| Day | Time Point | Parameter |
|--------------|----------------------|---------------|
| Screening | | HR, BP, RR, T |
| Day -1 | Check-in | HR, BP, RR, T |
| Day 1 | Predose | HR, BP, RR, T |
| Day 1 | Hour 2, Hour 4 | HR, BP, RR |
| Day 2 | | HR, BP, RR |
| Day 3 | | HR, BP, RR |
| Day 4 | | HR, BP, RR |
| Day 5 | | HR, BP, RR |
| Day 6 | | HR, BP, RR |
| Day 7 | | HR, BP, RR |
| Day 8 | EOT or ET* | HR, BP, RR, T |
| *performed a | t EOT or prior to ET | |

Descriptive statistics will be reported for vital sign measurements (blood pressure [BP], pulse [HR], and respiration rate [RR]) and change from baseline by cohort and time point. Baseline is the last non-missing predose measurement prior to dosing (Day 1 Predose), including unscheduled assessments. Postdose unscheduled values and ET results will not be used for calculation of descriptive statistics. All vital signs results will be listed by subject.

# 7.6 ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction])

Single 12-lead ECGs will be performed at the following time points:

**Table 7.6: ECG Time Points** 

Descriptive statistics will be reported for ECG parameters and change from baseline by cohort and time point. Baseline is the last non-missing predose measurement prior to dosing (Day -1), including unscheduled assessments. Postdose unscheduled values and ET results will not be used for calculation of descriptive statistics. All ECG interval parameters will be listed by subject and time point of collection with QTcF > 450 msec and change from baseline > 30 msec flagged.

# 7.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary, Version 01Sep2018 B3 and listed.

# 7.8 Physical Examination

A full physical examination will be performed at Screening and on Day 8 or upon ET. Abbreviated physical examinations will be performed at Check-in (Day -1) and 1 hour postdose. Symptom-driven physical examinations may be performed at other times, at the PI's or designee's discretion. Abnormal findings will be reported as medical history or adverse events by the clinical site. Physical examination results will be listed by subject and time point.

# 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

Paired t-tests to evaluate the effect of renal function group were added in the analysis plan.

The rest of the analyses described in this SAP are aligned with those analyses described in the protocol.

## 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.3 or higher.

# 9.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

# Section 10:

Table 10-1 Summary of Disposition (Safety Population)

#### Section 11:

Table 11-1 Demographic Summary (Safety Population)

## **Total Plasma LOXO-292**

Table 11-2 Summary of Total Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to

Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

- Table 11-3 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment
  Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)
- Table 11-4 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Moderate Renal
  Impairment Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)
- Table 11-5 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment
  Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)
- Table 11-6 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment
  Versus Healthy Matched Control Subjects (Pharmacokinetic
  Population)
- Table 11-7 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Moderate Renal
  Impairment Versus Healthy Matched Control Subjects
  (Pharmacokinetic Population)
- Table 11-8 Summary of Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment
  Versus Healthy Matched Control Subjects (Pharmacokinetic
  Population)
- Figure 11-1 Arithmetic Mean Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

- Figure 11-2 Individual Total Plasma LOXO-292 AUC0-t Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Figure 11-3 Individual Total Plasma LOXO-292 AUC0-inf Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Figure 11-4 Individual Total Plasma LOXO-292 Cmax Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

## **Unbound Plasma LOXO-292**

- Table 11-9 Summary of Unbound Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Table 11-10 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment
  Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)
- Table 11-11 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Moderate Renal
  Impairment Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)
- Table 11-12 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment
  Versus Healthy Matched Control Subjects (Paired T-Test)
  (Pharmacokinetic Population)

- Table 11-13 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment
  Versus Healthy Matched Control Subjects (Pharmacokinetic
  Population)
- Table 11-14 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Moderate Renal
  Impairment Versus Healthy Matched Control Subjects
  (Pharmacokinetic Population)
- Table 11-15 Summary of Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a Single
  Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment
  Versus Healthy Matched Control Subjects (Pharmacokinetic
  Population)
- Figure 11-5 Arithmetic Mean Unbound Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Figure 11-6 Individual Unbound Plasma LOXO-292 AUC0-t,u Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Figure 11-7 Individual Unbound Plasma LOXO-292 AUC0-inf,u Values,
  Geometric Means With Corresponding 95% CIs, and GMR With
  Corresponding 90% CIs Following Administration of a Single Dose of
  160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe
  Renal Impairment and to Healthy Matched Control Subjects
  (Pharmacokinetic Population)
- Figure 11-8 Individual Unbound Plasma LOXO-292 Cmax,u Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

## **Urine LOXO-292**

- Table 11-16 Summary of Urine LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)
- Figure 11-9 Arithmetic Mean Cumulative % Dose of LOXO-292 Excreted Unchanged in Urine Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

#### Section 12:

Table 12-1 Treatment-Emergent Adverse Event Frequency by Cohort – Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

# 9.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

## 14.1 Demographic Data Summary Tables

## 14.1.1 Demographic Tables

- Table 14.1.1.1 Summary of Disposition (Safety Population)
- Table 14.1.1.2 Demographic Summary (Safety Population)

## 14.2 Pharmacokinetic Data Summary Tables and Figures

## 14.2.1 Total Plasma LOXO-292 Tables

- Table 14.2.1.1 Total Plasma LOXO-292 Concentrations (ng/mL)
  Following Administration of a Single Dose of 160 mg
  LOXO-292 to Subjects with Mild Renal Impairment
  (Pharmacokinetic Population)
- Table 14.2.1.2 Total Plasma LOXO-292 Concentrations (ng/mL)
  Following Administration of a Single Dose of 160 mg
  LOXO-292 to Subjects with Moderate Renal Impairment
  (Pharmacokinetic Population)

| Table 14.2.1.3 | Total Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment (Pharmacokinetic Population) |
|---|---|
| Table 14.2.1.4 | Total Plasma LOXO-292 Concentrations (ng/mL)<br>Following Administration of a Single Dose of 160 mg<br>LOXO-292 to Healthy Matched Control Subjects<br>(Pharmacokinetic Population) |
| Table 14.2.1.5 | Total Plasma LOXO-292 Pharmacokinetic Parameters<br>Following Administration of a Single Dose of 160 mg<br>LOXO-292 to Subjects with Mild Renal Impairment<br>(Pharmacokinetic Population) |
| Table 14.2.1.6 | Total Plasma LOXO-292 Pharmacokinetic Parameters<br>Following Administration of a Single Dose of 160 mg<br>LOXO-292 to Subjects with Moderate Renal Impairment<br>(Pharmacokinetic Population) |
| Table 14.2.1.7 | Total Plasma LOXO-292 Pharmacokinetic Parameters<br>Following Administration of a Single Dose of 160 mg<br>LOXO-292 to Subjects with Severe Renal Impairment<br>(Pharmacokinetic Population) |
| Table 14.2.1.8 | Total Plasma LOXO-292 Pharmacokinetic Parameters<br>Following Administration of a Single Dose of 160 mg<br>LOXO-292 to Healthy Matched Control Subjects<br>(Pharmacokinetic Population) |
| Table 14.2.1.9 | Intervals (Hours) Used for Determination of Total Plasma<br>LOXO-292 Kel Values Following Administration of a<br>Single Dose of 160 mg LOXO-292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |
| Table 14.2.1.10 | Statistical Comparisons of Total Plasma LOXO-292<br>Pharmacokinetic Parameters Following Administration of a<br>Single Dose of 160 mg LOXO 292 to Subjects with Mild<br>Renal Impairment Versus Healthy Matched Control<br>Subjects (Paired T-Test) (Pharmacokinetic Population) |
| Table 14.2.1.11 | Statistical Comparisons of Total Plasma LOXO-292<br>Pharmacokinetic Parameters Following Administration of a<br>Single Dose of 160 mg LOXO 292 to Subjects with<br>Moderate Renal Impairment Versus Healthy Matched |

Control Subjects (Paired T-Test) (Pharmacokinetic Population)

- Table 14.2.1.12 Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Severe
  Renal Impairment Versus Healthy Matched Control
  Subjects (Paired T-Test) (Pharmacokinetic Population)
- Table 14.2.1.13 Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Mild
  Renal Impairment Versus Healthy Matched Control
  Subjects (Pharmacokinetic Population)
- Table 14.2.1.14 Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with
  Moderate Renal Impairment Versus Healthy Matched
  Control Subjects (Pharmacokinetic Population)
- Table 14.2.1.15 Statistical Comparisons of Total Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Severe
  Renal Impairment Versus Healthy Matched Control
  Subjects (Pharmacokinetic Population)

# 14.2.2 Total Plasma LOXO-292 Figures

- Figure 14.2.2.1 Mean (SD) Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.2.2 Mean Total Plasma LOXO-292 Concentration-Time
  Profiles Following Administration of a Single Dose of
  160 mg LOXO-292 to Subjects with Mild, Moderate, and
  Severe Renal Impairment and to Healthy Matched Control
  Subjects (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.2.3 Mean Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Semi-Log Scale) (Pharmacokinetic Population)

| Figure 14.2.2.4 | Individual Total Plasma LOXO-292 AUC0-t Values,<br>Geometric Means With Corresponding 95% CIs, and GMR<br>With Corresponding 90% CIs Following Administration of<br>a Single Dose of 160 mg LOXO-292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |
|---|---|
| Figure 14.2.2.5 | Individual Total Plasma LOXO-292 AUC0-inf Values,<br>Geometric Means With Corresponding 95% CIs, and GMR<br>With Corresponding 90% CIs Following Administration of<br>a Single Dose of 160 mg LOXO-292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |
| Figure 14.2.2.6 | Individual Total Plasma LOXO-292 Cmax Values,<br>Geometric Means With Corresponding 95% CIs, and GMR<br>With Corresponding 90% CIs Following Administration of<br>a Single Dose of 160 mg LOXO-292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |

# Note:

- Figures 14.2.2.4-6 are plots of AUCs and Cmax versus the cohorts.
- The x-axis will be the renal function and the y-axis will be the individual plasma PK parameters.

| Figure 14.2.2.7 | Scatter/Regression Plot of Individual Plasma LOXO-292<br>AUC0-t Versus eGFR |
|---|---|
| Figure 14.2.2.8 | Scatter/Regression Plot of Individual Plasma LOXO-292<br>AUC0-inf Versus eGFR |
| Figure 14.2.2.9 | Scatter/Regression Plot of Individual Plasma LOXO-292<br>Cmax Versus eGFR |

## Note:

- Figures 14.2.2.7-9 are scatter plots with regression lines.
- The x-axis will be the individual eGFR values and the y-axis will be the individual plasma PK parameters
- Figure 14.2.2.10 Scatter/Regression Plot of Individual Plasma LOXO-292 AUC0-t Versus CLcr
- Figure 14.2.2.11 Scatter/Regression Plot of Individual Plasma LOXO-292 AUC0-inf Versus CLcr

Figure 14.2.2.12 Scatter/Regression Plot of Individual Plasma LOXO-292 Cmax Versus CLcr

#### Note:

- Figures 14.2.2.10-12 are scatter plots with regression lines.
- The x-axis will be the individual CLcr values (found in the RFA dataset) and the y-axis will be the individual CLcr values

#### 14.2.3 Unbound Plasma LOXO-292 Tables

- Table 14.2.3.1 Concentrations of LOXO-292 (LOXO-292) (ng/mL), and Concentrations in the Buffer Chamber (LOXO-292 BC), Concentrations in the Plasma Chamber (LOXO-292 PC), % Recovery, and Fraction Unbound Obtained Following the Plasma Protein Binding Assay in Subjects with Mild Renal Impairment (Pharmacokinetic Population)
- Table 14.2.3.2 Concentrations of LOXO-292 (LOXO-292) (ng/mL), and Concentrations in the Buffer Chamber (LOXO-292 BC), Concentrations in the Plasma Chamber (LOXO-292 PC), % Recovery, and Fraction Unbound Obtained Following the Plasma Protein Binding Assay in Subjects with Moderate Renal Impairment (Pharmacokinetic Population)
- Table 14.2.3.3 Concentrations of LOXO-292 (LOXO-292) (ng/mL), and Concentrations in the Buffer Chamber (LOXO-292 BC), Concentrations in the Plasma Chamber (LOXO-292 PC), % Recovery, and Fraction Unbound Obtained Following the Plasma Protein Binding Assay in Subjects with Severe Renal Impairment (Pharmacokinetic Population)
- Table 14.2.3.4 Concentrations of LOXO-292 (LOXO-292) (ng/mL), and Concentrations in the Buffer Chamber (LOXO-292 BC), Concentrations in the Plasma Chamber (LOXO-292 PC), % Recovery, and Fraction Unbound Obtained Following the Plasma Protein Binding Assay in Healthy Matched Control Subjects (Pharmacokinetic Population)
- Table 14.2.3.5 Unbound Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| Table 14.2.3.6 | Unbound Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Moderate Renal Impairment (Pharmacokinetic Population) |
|---|---|
| Table 14.2.3.7 | Unbound Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment (Pharmacokinetic Population) |
| Table 14.2.3.8 | Unbound Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Healthy Matched Control Subjects (Pharmacokinetic Population) |
| Table 14.2.3.9 | Unbound Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population) |
| Table 14.2.3.10 | Unbound Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Moderate Renal Impairment (Pharmacokinetic Population) |
| Table 14.2.3.11 | Unbound Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment (Pharmacokinetic Population) |
| Table 14.2.3.12 | Unbound Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Healthy Matched Control Subjects (Pharmacokinetic Population) |
| Table 14.2.3.13 | Intervals (Hours) Used for Determination of Unbound Plasma LOXO-292 Kel Values Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population) |
| Table 14.2.3.14 | Statistical Comparisons of Unbound Plasma LOXO-292<br>Pharmacokinetic Parameters Following Administration of a<br>Single Dose of 160 mg LOXO 292 to Subjects with Mild |

Renal Impairment Versus Healthy Matched Control Subjects (Paired T-Test) (Pharmacokinetic Population)

- Table 14.2.3.15 Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with
  Moderate Renal Impairment Versus Healthy Matched
  Control Subjects (Paired T-Test) (Pharmacokinetic
  Population)
- Table 14.2.3.16 Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Severe
  Renal Impairment Versus Healthy Matched Control
  Subjects (Paired T-Test) (Pharmacokinetic Population)
- Table 14.2.3.17 Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Mild
  Renal Impairment Versus Healthy Matched Control
  Subjects (Pharmacokinetic Population)
- Table 14.2.3.18 Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with
  Moderate Renal Impairment Versus Healthy Matched
  Control Subjects (Pharmacokinetic Population)
- Table 14.2.3.19 Statistical Comparisons of Unbound Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of a
  Single Dose of 160 mg LOXO 292 to Subjects with Severe
  Renal Impairment Versus Healthy Matched Control
  Subjects (Pharmacokinetic Population)

# 14.2.4 Unbound Plasma LOXO-292 Figures

Figure 14.2.4.1 Mean (SD) Unbound Plasma LOXO-292 Concentration— Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Linear Scale) (Pharmacokinetic Population)
| Figure 14.2.4.2 | Mean Unbound Plasma LOXO-292 Concentration-Time<br>Profiles Following Administration of a Single Dose of<br>160 mg LOXO-292 to Subjects with Mild, Moderate, and<br>Severe Renal Impairment and to Healthy Matched Control<br>Subjects (Linear Scale) (Pharmacokinetic Population) |
|---|---|
| Figure 14.2.4.3 | Mean Unbound Plasma LOXO-292 Concentration-Time<br>Profiles Following Administration of a Single Dose of<br>160 mg LOXO-292 to Subjects with Mild, Moderate, and<br>Severe Renal Impairment and to Healthy Matched Control<br>Subjects (Semi-Log Scale) (Pharmacokinetic Population) |
| Figure 14.2.4.4 | Individual Unbound Plasma LOXO-292 AUC0-t,u Values,<br>Geometric Means With Corresponding 95% CIs, and GMR<br>With Corresponding 90% CIs Following Administration of<br>a Single Dose of 160 mg LOXO 292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |
| Figure 14.2.4.5 | Individual Unbound Plasma LOXO-292 AUC0-inf,u<br>Values, Geometric Means With Corresponding 95% CIs,<br>and GMR With Corresponding 90% CIs Following<br>Administration of a Single Dose of 160 mg LOXO 292 to<br>Subjects with Mild, Moderate, and Severe Renal<br>Impairment and to Healthy Matched Control Subjects<br>(Pharmacokinetic Population) |
| Figure 14.2.4.6 | Individual Unbound Plasma LOXO-292 Cmax,u Values,<br>Geometric Means With Corresponding 95% CIs, and GMR<br>With Corresponding 90% CIs Following Administration of<br>a Single Dose of 160 mg LOXO 292 to Subjects with Mild,<br>Moderate, and Severe Renal Impairment and to Healthy<br>Matched Control Subjects (Pharmacokinetic Population) |
| Note: | |
| • Figures 1 | 4.2.4.4-6 are plot of AUCs and Cmax versus the cohorts. |
| | is will be the renal function and the y-axis will be the l unbound plasma PK parameters. |
| Figure 14.2.4.7 | Scatter/Regression Plot of Individual Unbound Plasma<br>LOXO-292 AUC0-t,u Versus eGFR |

Scatter/Regression Plot of Individual Unbound Plasma

Scatter/Regression Plot of Individual Unbound Plasma

LOXO-292 AUC0-inf,u Versus eGFR

LOXO-292 Cmax,u Versus eGFR

Figure 14.2.4.8

Figure 14.2.4.9

#### Note:

- Figures 14.2.4.7-9 are scatter plots with regression lines.
- The x-axis will be the individual eGFR values (found in the RFA dataset) and the y-axis will be the individual unbound plasma PK parameters
- Figure 14.2.4.10 Scatter/Regression Plot of Individual Unbound Plasma LOXO-292 AUC0-t,u Versus CLcr

  Figure 14.2.4.11 Scatter/Regression Plot of Individual Unbound Plasma LOXO-292 AUC0-inf,u Versus CLcr
- Figure 14.2.4.12 Scatter/Regression Plot of Individual Unbound Plasma LOXO-292 Cmax,u Versus CLcr

#### Note:

- Figures 14.2.4.10-12 are scatter plots with regression lines.
- The x-axis will be the individual CLcr values (found in the RFA dataset) and the y-axis will be the individual unbound plasma PK parameters

#### 14.2.5 Urine LOXO-292 Tables

- Table 14.2.5.1 Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)
- Table 14.2.5.2 Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Moderate Renal Impairment (Pharmacokinetic Population)
- Table 14.2.5.3 Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment (Pharmacokinetic Population)
- Table 14.2.5.4 Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Healthy
  Matched Control Subjects (Pharmacokinetic Population)
- Table 14.2.5.5 Pharmacokinetic Parameters for Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| Table 14.2.5.6 | Pharmacokinetic Parameters for Urinary Excretion of |
|----------------|-------------------------------------------------------|
| | LOXO-292 Following Administration of a Single Dose of |
| | 160 mg LOXO-292 to Subjects with Moderate Renal |
| | Impairment (Pharmacokinetic Population) |

- Table 14.2.5.7 Pharmacokinetic Parameters for Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Severe Renal Impairment (Pharmacokinetic Population)
- Table 14.2.5.8 Pharmacokinetic Parameters for Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Healthy Matched Control Subjects (Pharmacokinetic Population)

## 14.2.6 Urine LOXO-292 Figures

- Figure 14.2.6.1 Arithmetic Mean (SD) Cumulative Amount of LOXO-292
  Excreted Unchanged in Urine Following Administration of
  a Single Dose of 160 mg LOXO-292 to Subjects with Mild,
  Moderate, and Severe Renal Impairment and to Healthy
  Matched Control Subjects (Linear Scale) (Pharmacokinetic
  Population)
- Figure 14.2.6.2 Arithmetic Mean Cumulative Amount of LOXO-292
  Excreted Unchanged in Urine Following Administration of
  a Single Dose of 160 mg LOXO-292 to Subjects with Mild,
  Moderate, and Severe Renal Impairment and to Healthy
  Matched Control Subjects (Linear Scale) (Pharmacokinetic
  Population)
- Figure 14.2.6.3 Arithmetic Mean (SD) Cumulative % Dose of LOXO-292 Excreted Unchanged in Urine Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.6.4 Arithmetic Mean Cumulative % Dose of LOXO-292

  Excreted Unchanged in Urine Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Linear Scale) (Pharmacokinetic Population)

#### 14.3 Safety Data Summary Tables

## 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Cohort Number of Subjects Reporting Events (% of Subject Dosed) (Safety Population)
- Table 14.3.1.2 Treatment-emergent Adverse Event Frequency by Cohort Number of Adverse Events (% of Total Adverse Events) (Safety Population)
- Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by Cohort, Severity Grade, and Relationship to Study Drug - Number of Subjects Reporting Events (Safety Population)
- Table 14.3.1.4 Treatment-Emergent Adverse Event Frequency by Cohort, Severity Grade, and Relationship to Study Drug - Number of Adverse Events (Safety Population)

# 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)

Note: If no serious adverse event occurred, a statement 'There was no serious adverse event recorded during the study.' will be added.

# 14.3.3. Narratives of Deaths, other Serious and Certain other Significant Adverse Events

#### 14.3.4. Abnormal Laboratory Value Listing (by Subject)

- Table 14.3.4.1 Out-of-Range Values and Unscheduled Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Unscheduled Results Hematology and Coagulation
- Table 14.3.4.3 Out-of-Range Values and Unscheduled Results Urinalysis
- Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

# 14.3.5. Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary Serum Chemistry (Safety Population)
- Table 14.3.5.2 Clinical Laboratory Change from Baseline Serum Chemistry (Safety Population)
- Table 14.3.5.3 Clinical Laboratory Shift from Baseline Serum Chemistry (Safety Population)

| Table 14.3.5.4 | Clinical Laboratory Summary – Hematology and Coagulation (Safety Population) |
|---|---|
| Table 14.3.5.5 | Clinical Laboratory Change from Baseline – Hematology and Coagulation (Safety Population) |
| Table 14.3.5.6 | Clinical Laboratory Shift from Baseline – Hematology and Coagulation (Safety Population) |
| Table 14.3.5.7 | Clinical Laboratory Summary – Urinalysis (Safety Population) |
| Table 14.3.5.8 | Clinical Laboratory Change from Baseline – Urinalysis (Safety Population) |
| Table 14.3.5.9 | Clinical Laboratory Shift from Baseline – Urinalysis (Safety Population) |
| Table 14.3.5.10 | Vital Sign Summary (Safety Population) |
| Table 14.3.5.11 | Vital Sign Change from Baseline (Safety Population) |
| Table 14.3.5.12 | 12-Lead Electrocardiogram Summary (Safety Population) |
| Table 14.3.5.13 | 12-Lead Electrocardiogram Change from Baseline (Safety Population) |

## 9.3 Section 16 Data Listings

Note: Virology test results (Hepatitis and HIV) that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in the database transfer. The date of sample collection only will be provided in the database and listings.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

### **16.1** Study Information

| Appendix 16.1.9 | Statistical Methods |
|---|---|
| Appendix 16.1.7.2 | Healthy Control Subjects Matched to Renal Function Groups |
| Appendix 16.1.10.1 | Clinical Laboratory Reference Ranges |

### 16.2. Subject Data Listings

### 16.2.1. Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (Safety Population)

#### 16.2.2. Protocol Deviations

# Appendix 16.2.2 Protocol Deviations

Note: Protocol deviations will be provided by the clinical study manager as Microsoft Excel file and read into the SDTM to generate the data listing.

# 16.2.3. Subjects Excluded from Pharmacokinetic Analysis

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic Analysis Note: Appendix 16.2.3 will be generated in MS Word for inclusion in the CSR.

# 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|-------------------|--------------------------------------------------|
| Appendix 16.2.4.2 | Physical Examination (Safety Population) |
| Appendix 16.2.4.3 | Medical and Surgical History (Safety Population) |
| Appendix 16.2.4.4 | Assessment of Renal Function (Safety Population) |

# 16.2.5. Compliance and Drug Concentration Data

| Appendix 16.2.5.1 | Subject Eligibility (Safety Population) |
|---|---|
| Appendix 16.2.5.2 | Test Compound Administration Times (Safety Population) |
| Appendix 16.2.5.3 | PK Blood Draw Times and Protein Binding (Safety Population) |
| Appendix 16.2.5.4 | Urine Collection Times (Safety Population) |
| Appendix 16.2.5.5 | Follow-Up Phone Call (Safety Population) |
| Appendix 16.2.5.6 | Prior and Concomitant Medications (Safety Population) |

# 16.2.6 Individual Pharmacokinetic Response Data

| Appendix 16.2.6.1 | Individual Total and Unbound Plasma LOXO-292<br>Concentrations Versus Time Profiles Following<br>Administration of a Single Dose of 160 mg LOXO-292<br>to Subject <#> (Linear and Semi-Log Scale) |
|---|---|
| Appendix 16.2.6.2 | Individual Cumulative Amount of LOXO-292 Excreted Unchanged in Urine Following Administration of a Single Dose of 160 mg LOXO-292 to Subject <#> (Linear Scale) |
| Appendix 16.2.6.3 | Individual Cumulative % Dose of LOXO-292 Excreted Unchanged in Urine Following Administration of a Single Dose of 160 mg LOXO-292 to Subject <#> (Linear Scale) |

## **16.2.7** Adverse Events Listings

| Appendix 16.2.7.1 | Adverse Events (I of II) (Safety Population) |
|-------------------|-----------------------------------------------------|
| Appendix 16.2.7.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.3 | Adverse Event Comments (Safety Population) |
| Appendix 16.2.7.4 | Adverse Event Preferred Term Classification (Safety |
| | Population) |

# 16.2.8 Listings of Individual Laboratory Measurements and Other Safety Observations

- Appendix 16.2.8.1.1.1 Clinical Laboratory Report Serum Chemistry (Conventional Units) (Safety Population)
- Appendix 16.2.8.1.1.2 Clinical Laboratory Report Serum Chemistry (SI Units) (Safety Population)
- Appendix 16.2.8.1.2.1 Clinical Laboratory Report Hematology and Coagulation (Conventional Units) (Safety Population)
- Appendix 16.2.8.1.2.2 Clinical Laboratory Report Hematology and Coagulation (SI Units) (Safety Population)
- Appendix 16.2.8.1.3.1 Clinical Laboratory Report Urinalysis (Conventional Units) (Safety Population)
- Appendix 16.2.8.1.3.2 Clinical Laboratory Report Urinalysis (SI Units) (Safety Population)
- Appendix 16.2.8.1.4.1 Clinical Laboratory Report Serum FSH (Conventional Units) (Safety Population)
- Appendix 16.2.8.1.4.2 Clinical Laboratory Report Serum FSH (SI Units) (Safety Population)
- Appendix 16.2.8.1.5 Clinical Laboratory Report Urine Drug Screening (Safety Population)
- Appendix 16.2.8.1.6 Clinical Laboratory Report Comments (Safety Population)
- Appendix 16.2.8.1.7 Clinical Laboratory Serology Samples (Safety Population)
- Appendix 16.2.8.2 Vital Signs (Safety Population)
- Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

### 10. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables and figures that will be presented and included in the final CSR. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 8 and post-text tables in Courier New size font 9. These tables will be generated according to the ADaM Model 2.1 and ADaM implementation guide 1.1.

# 10.1 In-text Table Shells

**Table 10-1 Summary of Disposition (Safety Population)** 

| Disposition | Subjects with<br>Mild RI | Subjects with<br>Moderate RI | Subjects with<br>Severe RI | Healthy Matched<br>Control Subjects | Overall |
|---|---|---|---|---|---|
| Enrolled | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Completed Study | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Discontinued Early | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason1></reason1> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason2></reason2> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

RI = Renal impairment

Source: Table 14.1.1.1

DDMMMYYYY HH:MM

**Table 11-1 Demographic Summary (Safety Population)** 

| Trait | | Subjects with<br>Mild RI | Subjects with<br>Moderate RI | Subjects with<br>Severe RI | Healthy Matched<br>Control Subjects | Overall |
|---|---|---|---|---|---|---|
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African<br>American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yr) | n | XX | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Height (cm) | n | XX | XX | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XXX | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Maximum | XXX | XXX | XXX | XXX | XXX |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

BMI = Body mass index

Source: Table 14.1.1.2

DDMMMYYYY HH:MM

**Programmer Note:** Weight (kg) and BMI (kg/m²) will also be summarized in the table above. Weight, height, and BMI will be summarized at Screening.

RI = Renal impairment

<sup>\*</sup> Age is calculated from the date of dosing.

In-text Tables 11-2, 11-9, and 11-16 will be in the following format:

Table 11-2 Summary of Total Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

| | | | | Healthy Matched Control |
|---|---|---|---|---|
| Pharmacokinetic Parameters | Subjects with Mild RI | Subjects with Moderate RI | Subjects with Severe RI | Subjects |
| Param1 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

RI = Renal impairment

AUCs and Cmax values are presented as geometric mean (geometric CV%).

Tmax values are presented as median (min, max).

Other parameters are presented as arithmetic mean ( $\pm$  SD).

Source: Tables 14.2.1.5 to 14.2.1.8

# **Notes for Generating the Actual Table:**

Presentation of Data:

- The following PK parameters will be presented in the following order:
  - o Table 11-2 (plasma): AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, t1/2, CL/F, and Vz/F
    - Source: Tables 14.2.1.5 to 14.2.1.8
  - o Table 11-9 (unbound plasma): AUC0-t,u, AUC0-inf,u, Cmax,u, CL/F,u, and Vz/F,u
    - Source: Tables 14.2.3.9 to 14.2.3.12
  - o Table 11-16 (urine): Ae0-t, CLr, and Fe
    - Source: Tables 14.2.5.5 to 14.2.5.8
- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells



In-text Tables 11-3 to 11-5 and 11-10 to 11-12 will be in the following format:

Table 11-3 Summary of Statistical Comparisons of Total Plasma LOXO-292
Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg
LOXO-292 to Subjects with Mild Renal Impairment Versus Corresponding Healthy Matched
Control Subjects (Paired T-Test) (Pharmacokinetic Population)

| | n | GMR (%) | 90% Confidence Interval | p-value |
|----------------|----|---------|-------------------------|---------|
| Parameter | | W 10 | | |
| param1 (units) | XX | XX.XX | XX.XX - XX.XX | X.XXXX |
| param2 (units) | XX | XX.XX | XX.XX - XX.XX | X.XXXX |
| param3 (units) | XX | XX.XX | XX.XX - XX.XX | X.XXXX |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Parameters were In-transformed prior to analysis and n is the number of paired differences (i.e, RI - Healthy).

Geometric Mean Ratio (GMR) and 90% confidence intervals (CIs) are calculated by exponentiating the mean difference (RI – healthy) and the associated 90 % confidence intervals derived from the paired t-test and multiplying by 100.

Source: Table 14.2.1.10

### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- The following PK parameters will be presented in the following order:
  - o Table 11-3 through 11-5: AUC0-t, AUC0-inf, and Cmax
  - o Table 11-10 through 11-12: AUC0-t,u, AUC0-inf,u, and Cmax,u
- n will be presented as an integer (with no decimal);
- All statistics will be presented with same precision as defined in post-text shells
- Source:
  - o Table 11-3: Table 14.2.1.10
  - o Table 11-4: Table 14.2.1.11
  - o Table 11-5: Table 14.2.1.12
  - o Table 11-10: Table 14.2.1.14
  - o Table 11-11: Table 14.2.1.15
  - o Table 11-12: Table 14.2.1.16



RI = Renal impairment

In-text Tables 11-6 to 11-8 and 11-13 to 11-15 will be in the following format:

Table 11-6 Summary of Statistical Comparisons of Total Plasma LOXO-292
Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg
LOXO-292 to Subjects with Mild Renal Impairment Versus Healthy Matched Control
Subjects (Pharmacokinetic Population)

| | Subjects with Mild | RI (Test) | Healthy Matched Con-<br>Subjects (Reference | 1000000000 | GMR (%) | 90% Confidence Interval |
|---|---|---|---|---|---|---|
| Parameter | Geometric LSMs | n | Geometric LSMs | n | | |
| param1 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX |
| param2 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX |
| param3 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

RI = Renal impairment

Parameters were In-transformed prior to analysis.

Geometric least-squares means (LSMs) are calculated by exponentiating the LSMs derived from the ANCOVA.

Geometric Mean Ratio (GMR) = 100\*(test/reference)

Source: Table 14.2.1.13

# **Notes for Generating the Actual Table:**

Presentation of Data:

- The following PK parameters will be presented in the following order:
  - o Table 11-3 through 11-5: AUC0-t, AUC0-inf, and Cmax
  - o Table 11-13 through 11-5: AUC0-t,u, AUC0-inf,u, and Cmax,u
- n will be presented as an integer (with no decimal);
- All statistics will be presented with same precision as defined in post-text shells
- Source:
  - o Table 11-3: Table 14.2.1.13
  - o Table 11-4: Table 14.2.1.14
  - o Table 11-5: Table 14.2.1.15
  - o Table 11-13: Table 14.2.1.17
  - o Table 11-14: Table 14.2.1.18
  - o Table 11-15: Table 14.2.1.19



Table 12-1 Treatment-Emergent Adverse Event Frequency by Cohort –
Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

| Adverse Events* | Subjects with<br>Mild RI | Subjects with<br>Moderate RI s | Subjects with<br>Severe RI | Healthy Matched<br>Control Subjects | Overall |
|---|---|---|---|---|---|
| Number of Subjects Dosed | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects Without TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| System Organ Class 1 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Preferred Term 1 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Preferred Term 2 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| System Organ Class 2 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Preferred Term 1 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Preferred Term 2 | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Although a subject may have had 2 or more clinical adverse experiences, the subject is counted only once within a category. The same subject may appear in different categories.

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity.

Source: Table 14.3.1.1

DDMMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

RI = Renal impairment

<sup>\*</sup> Adverse events are coded using MedDRA® Version 21.1 by System Organ Class and Preferred Term.

TEAE = Treatment-emergent Adverse event

# 10.2 Figures Shells

In-text Figures 11-1, 11-5, and 11-9, Figures 14.2.2.2, 14.2.4.2, 14.2.6.2, and 14.2.6.4 will be in the following format:

Figure 11-1 Arithmetic Mean Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)



Statistical Analysis Plan, 23 May 2019


# **Notes for Generating the Actual Mean Figure:**

- Figures 11-1 and 14.2.2.2:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Total Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Figures 11-5 and 14.2.4.2:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Unbound Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Figures 11-9 and 14.2.6.4:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - Y-axis label will be "Cumulative % Dose of LOXO-292 Excreted Unchanged (%)"
  - o X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886

- Figure 14.2.6.2:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Cumulative Amount of LOXO-292 Excreted Unchanged (ng)"
  - o X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.



Figures 14.2.2.1, 14.2.4.1, 14.2.6.1, and 14.2.6.3 will be in the following format:

Figure 14.2.2.1 Mean (SD) Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Linear Scale) (Pharmacokinetic Population)



## **Notes for Generating the Actual Mean Figure:**

- Figure 14.2.2.1:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Total Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Figure 14.2.4.1:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Unbound Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Figure 14.2.6.1:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - Y-axis label will be "Cumulative Amount of LOXO-292 Excreted Unchanged (ng)"
  - o X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886

- Figure 14.2.6.3:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Cumulative % Dose of LOXO-292 Excreted Unchanged (%)"
  - o X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.



Figures 14.2.2.3 and 14.2.4.3 will be in the following format:

Figure 14.2.2.3 Mean Total Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Semi-Log Scale) (Pharmacokinetic Population)



# **Notes for Generating the Actual Mean Figure:**

- Figure 14.2.2.3:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Total Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Figure 14.2.4.3:
  - o Legend will be:
    - Subjects with Mild RI (n = X)
    - Subjects with Moderate RI (n = X)
    - Subjects with Severe RI (n = X)
    - Healthy Matched Control Subjects (n = X)
  - o Y-axis label will be "Unbound Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.



In-text Figures 11-2 through 11-4, 11-6 through 11-8, and Figures 14.2.2.4 through 14.2.2.6 and 14.2.4.4 through 14.2.4.6 will be in the following format:

Figure 11-2 Individual Total Plasma LOXO-292 AUC0-t Values, Geometric Means With Corresponding 95% CIs, and GMR With Corresponding 90% CIs Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)



800 mg (A)/400 mg (B) GMR 90% CI: XX.XX [XX.XX, XX.XX]

# **Notes for Generating the Actual Figure:**

- The individual values by cohort will be presented in an almost vertical plane, and only staggered if there are some overlaps of symbols. The geometric mean and 95% CI will accompany each cohort. The GMR and 90% CI for each comparison from the paired t-test will be inserted below the x-axis as a footnote.
- Use different symbols for each cohort
- Legend will be:
  - o Subjects with Mild RI (n = X)
  - O Subjects with Moderate RI (n = X)
  - O Subjects with Severe RI (n = X)
  - Healthy Matched Control Subjects (n = X)
- Y-axis label will be the PK parameter with the appropriate unit: AUC0-t, AUC0-t,u, AUC0-inf, AUC0-inf,u, Cmax, or Cmax,u
- X-axis label will be the cohorts: "Mild/Moderate/Severe/Healthy"

Appendices 16.2.6.1 through 16.2.6.3 will be in the following format:

Appendix 16.2.6.1
Individual Total and Unbound Plasma LOXO-292 Concentrations Versus Time Profiles
Following Administration of a Single Dose of 160 mg LOXO-292 to Subject <#> (Linear and Semi-Log Scale)



## **Notes for Generating the Actual Individual Figure:**

- Appendix 16.2.6.1:
  - o Legend will be one of the following:
    - Subjects with Mild RI
    - Subjects with Moderate RI
    - Subjects with Severe RI
    - Healthy Matched Control Subjects
  - Y-axis label will be "Total or Unbound Plasma LOXO-292 Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL.
- Appendix 16.2.6.2 (only linear scale presented):
  - Legend will be one of the following:
    - Subjects with Mild RI
    - Subjects with Moderate RI
    - Subjects with Severe RI
    - Healthy Matched Control Subjects
  - Y-axis label will be "Cumulative Amount of LOXO-292 Excreted Unchanged (ng)"
  - X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.
- Appendix 16.2.6.3 (only linear scale presented):
  - o Legend will be one of the following:
    - Subjects with Mild RI
    - Subjects with Moderate RI
    - Subjects with Severe RI
    - Healthy Matched Control Subjects
  - Y-axis label will be "Cumulative % Dose of LOXO-292 Excreted Unchanged (ng)"
  - X-axis label will be "Interval End (hr)"
  - o Add in footnote: LLOQ value for LOXO-292 in urine is 5.00 ng/mL.



#### 10.3 Post-text Table Shells

Page X of X

Table 14.1.1.1 Summary of Disposition (Safety Population)

| | | Cohort | | | |
|--------------------|------|----------|--------|---------|---------|
| Disposition | Mild | Moderate | Severe | Healthy | Overall |
| Enrolled | XX | XX | XX | XX | XX |
| Completed | XX | XX | XX | XX | XX |
| Discontinued Early | XX | XX | XX | XX | XX |
| Reason 1 | XX | XX | XX | XX | XX |
| Reason 2 | XX | XX | XX | XX | XX |
| Reason 3 | XX | XX | XX | XX | XX |
| etc. | | | | | |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions:

Mild: Subjects with mild renal impairment

Moderate: Subjects with moderate renal impairment Severe: Subjects with severe renal impairment Healthy: Healthy matched control subjects

CCI

DDMMMYYYY HH:MM


Table 14.1.1.2 Demographic Summary (Safety Population)

| | | | Cohort | | | |
|---|---|---|---|---|---|---|
| Trait | | Mild | Moderate | Severe | Healthy | Overall |
| Sex | Male<br>Female | X ( XX%)<br>X ( XX%) | X ( XX%)<br>X ( XX%) | | | X ( XX%)<br>X ( XX%) |
| Race | Asian<br>Black or African American<br>White | X ( XX%)<br>X ( XX%)<br>X ( XX%) | | X ( XX%) | X ( XX%) | X ( XX%)<br>X ( XX%)<br>X ( XX%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | X ( XX%)<br>X ( XX%) | | , , | , , | , , |
| Age*(yr) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.X<br>X.XX<br>XX<br>XX.X<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX.X<br>XX |
| Height (cm) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.X<br>X.XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X | XX<br>XX.X<br>X.XX<br>XX<br>XX.X<br>XX |

**Programmer Note:** Also include weight (kg) and BMI (kg/ $m^2$ ). Weight, height and BMI will be summarized at Screening. Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions:

Mild: Subjects with mild renal impairment

Moderate: Subjects with moderate renal impairment

Severe: Subjects with severe renal impairment

Healthy: Healthy matched control subjects

\* Age is calculated from the date of dosing.

BMI = Body mass index

DDMMYYYY HH:MM

Statistical Analysis Plan, 23 May 2019


# Tables 14.2.1.1 through 14.2.1.4, and 14.2.3.5 through 14.2.3.8 will be in the following format:

Table 14.2.1.1 Total Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| | | Sample Times (hr) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | | | | | | | | |
| Number | Predose | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 1.00 ng/mL are treated as 0 before the first quantifiable concentration and as missing elsewhere.

<sup>. =</sup> Value missing or not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Concentrations will be presented to same precision as in the bioanalytical data.
- Summary statistics presentation with respect to the precision of the bioanalytical data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

# Programmer Note:

- PK Time points are: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose.
- Tables 14.2.3.5 through 14.2.3.8: the unbound plasma LOXO-292 concentrations will be calculated by multiplying the
  measured LOXO-292 concentrations by the fraction of unbound LOXO-292 at each sampling time point for each subject. The
  fraction unbound will be calculated in Table 14.2.3.1 through 14.2.3.4.

Per study design needs, the following changes are made to this table relative to Celerion standard:

1. Please remove the "Treatment Sequence" and "Study Period" columns



DDMMMYYYY HH:MM DDMMMYYYY HH:MM DDMMMYYYY HH:MM

# Tables 14.2.1.5 through 14.2.1.8, and 14.2.3.9 through 14.2.3.12 will be in the following format:

Table 14.2.1.5 Total Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| | | | Param | neters | | |
|---|---|---|---|---|---|---|
| Subject | param1 | param2 | param3 | param4 | param5 | param6 |
| Number | (units) | (units) | (units) | (units) | (units) | (units) |
| XXX-XXX | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | X.XX | X.XX | XXX | XXX | XX.X | X.XXX |
| XXX-XXX | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| Median | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Maximum | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| Geom Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Geom CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| L95% CI (Geom Mean) | XX.X | XX.X | | XX.X | | |
| U95% CI (Geom Mean) | XX.X | XX.X | | XX.X | | |

<sup>. =</sup> Value missing or not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- The following PK parameters will be presented in the following order:
  - o Table 14.2.1.5 through 14.2.1.8: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, t1/2, CL/F, and Vz/F
  - o Table 14.2.3.9 through 14.2.3.12: AUC0-t,u, AUC0-inf,u, Cmax,u, CL/F,u, and Vz/F,u
- n will be presented as an integer (with no decimal);
- Parameter values for exposure-based parameters (i.e. AUCs, AUC%extrap, Cmax, CL/F, and Vz/F) will be presented with, at
  maximum, the precision of the bioanalytical data, and, at minimum, 3 significant figures (to be determined by the PKist once
  the bioanalytical data are received).
  - Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of significant figures.
- Values for time-based parameters (i.e. Tmax, and t½) will be presented with 2 decimals.
  - Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of decimals.
- Values for rate constants (i.e. Kel) will be presented with 3 significant figures.
  - Summary statistics for Kel will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of significant figures.
- CV% and Geom CV% for all parameters will be presented with 1 decimal
- 95% CI (Geom Mean) will be presented for AUC0-t, AUC0-inf and Cmax only
- 95% CI (Geom Mean) will be presented with 2 decimals
- Remove 'Treatment Sequence' and 'Study Period'



### Tables 14.2.1.9 and 14.2.3.13 will be in the following format:

Table 14.2.1.9 Intervals (Hours) Used for Determination of Total Plasma LOXO-292 Kel Values Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild, Moderate, and Severe Renal Impairment and to Healthy Matched Control Subjects (Pharmacokinetic Population)

| Subject<br>Number | Cohort | Interval | R2 | n |
|-------------------|--------|-------------|-------|---|
| XXX-XXX | Х | xx.x - xx.x | x.xxx | Х |
| XXX-XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | X | XX.X - XX.X | X.XXX | X |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions:

Mild: Subjects with mild renal impairment

Moderate: Subjects with moderate renal impairment Severe: Subjects with severe renal impairment Healthy: Healthy matched control subjects

R2 = Coefficient of determination

n = Number of points used in Kel calculation

. = Kel value not reportable.

# **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Interval start and stop times will be presented to 1 decimal or 3 significant figures minimum;
- R2 will be presented to 3 decimals;
- n will be presented as an integer (with no decimal)



### Tables 14.2.1.10 through 14.2.1.12 and 14.2.3.14 through 14.2.3.16 will be in the following format:

Table 14.2.1.10 Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment Versus Corresponding Healthy Matched Control Subjects (Paired t-test) (Pharmacokinetic Population)

| | | | Geometric Mean | 90% | |
|-----------|--------|----|----------------|----------------------|---------|
| Parameter | (unit) | n | Ratio (%) | Confidence Intervals | p-value |
| Param1 | (unit) | XX | XXX.XX | XXX.XX - XXX.XX | X.XXXX |
| Param2 | (unit) | XX | XXX.XX | XXX.XX - XXX.XX | X.XXXX |
| Param3 | (unit) | XX | XXX.XX | XXX.XX - XXX.XX | X.XXXX |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

RI = Renal impairment

Parameters were ln-transformed prior to analysis and n is the number of paired differences (i.e., RI - Healthy). Geometric Mean Ratio (GMR) and 90% confidence intervals (CIs) are calculated by exponentiating the mean difference (RI - healthy) and the associated 90% confidence intervals derived from the paired t-test and multiplying by 100

# **Notes for Generating the Actual Table:**

#### Presentation of Data:

- p-value will be presented with 4 decimals.
- Geometric Mean Ratio and 90% CI will be presented to 2 decimal places.
- PK parameters to be presented are
  - o Tables 14.2.1.10 through 14.2.1.12 : AUC0-t, AUC0-inf, and Cmax
  - o Tables 14.2.3.14 through 14.2.3.16 : AUC0-t,u AUC0-inf,u, and Cmax,u



#### Tables 14.2.1.13 through 14.2.1.15 and 14.2.3.17 through 14.2.3.19 will be in the following format:

Table 14.2.1.13 Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment Versus Healthy Matched Control Subjects (Pharmacokinetic Population)

| | | | Treatment Geometric LSMs | | tment | Geometric<br>Mean | 90% |
|---|---|---|---|---|---|---|---|
| Parameter | (unit) | Mild | (n) | Healthy | (n) | Ratio | Confidence Intervals |
| Param1 | (unit) | X.XX | (n) | X.XX | (n) | XXX.XX | XXX.XX - XXX.XX |
| Param2 | (unit) | X.XX | (n) | X.XX | (n) | XXX.XX | XXX.XX - XXX.XX |
| Param3 | (unit) | X.XX | (n) | X.XX | (n) | XXX.XX | xxx.xx - xxx.xx |

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions:

Mild: Subjects with mild renal impairment

Healthy: Healthy matched control subjects

Parameters were In-transformed prior to analysis.

Geometric least-squares means (LSMs) are calculated by exponentiating the LSMs from ANCOVA.

Geometric Mean Ratio is calculated by exponentiating the LSM difference (Renal impaired - healthy) and multiplying by 100.

## Notes for Generating the Actual Table:

#### Presentation of Data:

- Geometric LSMs will be presented to the same precision as the Mean in the PK parameter table.
- Geometric Mean Ratio and 90% CI will be presented to 2 decimal places.
- PK parameters to be presented are
  - o Tables 14.2.1.13 through 14.2.1.15 : AUC0-t, AUC0-inf, and Cmax
  - o Tables 14.2.3.17 through 14.2.3.19 : AUC0-t,u AUC0-inf,u, and Cmax,u


#### Tables 14.2.3.1 through 14.2.3.4 will be presented in the following format:

Table 14.2.3.1 Concentrations of LOXO-292 (LOXO-292) (ng/mL), and Concentrations in the Buffer Chamber (LOXO-292 BC), and Concentrations in the Plasma Chamber (LOXO-292 PC), % Recovery, and Fraction Unbound Obtained Following the Plasma Protein Binding Assay in Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| Number | LOXO-292 | | LOXO-292 PC | Recovery (%) | Fraction<br>Unbound |
|---|---|---|---|---|---|
| XXX-XXX | XXX | XX.X | XXX | XX.XX | X.XXX |
| XXX—XXX | XXX | XX.X | XXX | XX.XX | X.XXX |
| XXX-XXX | X | XX.X | XXX | XX.XX | X.XXX |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX |

LOXO-292: Total concentration, LOXO-292 concentration in matrix prior to dialysis

LOXO-292 BC: Buffer concentration, LOXO-292 concentration in the buffer chamber following dialysis

LOXO-292 PC: Plasma concentration, LOXO-292 concentration in the plasma chamber following dialysis

Recovery = (LOXO-292 BC + LOXO-292 PC) / LOXO-292

Fraction unbound = LOXO-292 BC / LOXO-292 PC

<sup>. =</sup> Value missing or not reportable.

### **Notes for Generating the Actual Table:**

Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Concentrations will be presented to same precision as in the bioanalytical data.
- Summary statistics presentation with respect to the precision of the bioanalytical data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal
- The 'Recovery' will be calculated as follow: (LOXO-292 BC + LOXO-292 PC) / LOXO-292
- The 'Fraction unbound' will be calculated as follow: LOXO-292 BC / LOXO-292 PC

### Tables 14.2.5.1 through 15.2.5.4 will be presented in the following format:


Table 14.2.5.1 Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

---- Parameters -----Predose t1 - t2 Hours t2-t3 Hours Subject Vol Aet1-t2 Vol Aet2-t3 Conc Conc Vol Conc Number (units) (units) (units) (units) (units) (units) (units) (unit) XXX-XXXX.XX X.XX XX.XX X.XX X.XX X.XX X.XX X.XX XXX-XXX X.XXX.XXXX.XX X.XX X.XX X.XX X.XX X.XX XX.XX XXX-XXX X.XXX.XX X.XX X.XX X.XX X.XX X.XX Χ Χ Χ Χ Χ Χ Χ Χ n X.XXX X.XXXXX.XXX X.XXXX.XXXX.XXX X.XXX X.XXXMean SD X.XXXX X.XXXX XX.XXX X.XXXX X.XXXX X.XXXXX.XXXXX.XXXXCV (%) X.XX.XXX.X Х.Х Х.Х Х.Х X.XХ.Х SEM X.XXXX X.XXXXXX.XXXX X.XXXXX.XXXX X.XXXXX.XXXXX.XXXXMinimum X.XXX.XXXX.XX X.XX X.XXX.XXX.XX X.XX Median X.XXX X.XXXXX.XXX X.XXXX.XXXX.XXXX.XXX X.XXXMaximum X.XXX.XX XX.XX X.XX X.XXX.XX X.XX X.XX

<sup>. =</sup> Value missing or not reportable.

For the calculation of summary statistics and urinary excretion parameters, concentration values that are BLQ of 5.00 ng/mL are treated as 0.

#### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Intervals are: predose, and 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours postdose
- Parameters to be presented:
  - o Predose: conc <unit> and volume <unit> only
  - o Each postdose interval: conc <unit>, volume <unit>, Aet1-t2 <unit>
- Concentrations will be presented to same precision as in the bioanalytical data. Volume will be presented to the same precision as the CRF.
  - Note: If the amount of urine excreted was captured in the CRF as urine weight (g), it will be converted to volume (mL) using the assumed density of 1 g/mL
  - o The units of Ae may be presented as mg if the overall cumulative value is more than 1 mg.
- Summary statistics presentation with respect to the precision of the bioanalytical data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

CCI

### Table 14.2.5.5 through 14.2.5.8 will be presented as follow:


Table 14.2.5.5 Pharmacokinetic Parameters for Urinary Excretion of LOXO-292 Following Administration of a Single Dose of 160 mg LOXO-292 to Subjects with Mild Renal Impairment (Pharmacokinetic Population)

| | | Parameters | |
|-----------|--------|------------|--------|
| Subject | Ae0-t | Fe | CLr |
| Number | (unit) | (%) | (unit) |
| XXX-XX | X.XX | X.XX | X.XX |
| XXX-XX | X.XX | X.XX | X.XX |
| XXX-XX | X.XX | X.XX | X.XX |
| n | X | X | X |
| Mean | X.XXX | X.XXX | X.XXX |
| SD | X.XXXX | X.XXXX | X.XXXX |
| CV% | X.X | X.X | Х.Х |
| SEM | X.XXXX | X.XXXX | X.XXXX |
| Minimum | X.XX | X.XX | X.XX |
| Median | X.XXX | X.XXX | X.XXX |
| Maximum | X.XX | X.XX | X.XX |
| Geom Mean | X.XXX | X.XXX | X.XXX |
| Geom CV% | X.X | х.х | X.X |

<sup>. =</sup> Value missing or not reportable.

For the calculation of summary statistics and urinary excretion parameters, concentration values that are BLQ of 5.00 ng/mL are treated as 0.

### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- PK parameters to present: Ae0-t <unit>, Fe <%>, CLr <unit>
  - Ae0-t is CumAe in Celerion standard programs, where t is the end time of the last interval with concentration data available
  - o Fe is CumFe in Celerion standard programs
- Ae0-t will be presented to the same precision as the bioanalytical data; Fe will be presented to 3 decimal places; CLr will be presented to 3 significant figures.
- Note: If the amount of urine excreted was captured in the CRF as urine weight (g), it will be converted to volume (mL) using the assumed density of 1 g/mL
- Summary statistics: n = integer; Mean, Median, and Geom Mean +1; SD and SEM +2; Min and Max +0; CV% and Geom CV% to 1 decimal

Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Cohort - Number of Subjects Reporting Events (% of Subject Dosed) (Safety Population)

| | Cohort | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | | ild | | derate | | evere | Healthy | | 70 | erall |
| Number of Subjects Dosed | Х | (100%) | X | (100%) | Х | (100%) | X | (100%) | Χ | (100%) |
| Number of Subjects with TE Adverse Events | Χ | (XX%) | X | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Number of Subjects without TE Adverse Events | Χ | (XX%) | Χ | (XX%) | Х | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Nervous system disorders | Х | (XX%) | Х | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) |
| Dizziness | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Headache | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Presyncope | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Respiratory, thoracic and mediastinal disorders | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Dry throat | Χ | (XX%) | X | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Oropharyngeal pain | Χ | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | Χ | (XX%) |
| Sinus congestion | Χ | (XX%) | X | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Sneezing | Χ | (XX%) | X | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| General disorders and administration site conditions | Χ | (XX%) | X | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Fatique | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) |
| Thirst | Χ | (XX%) | Χ | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| etc. | | | | | | | | | | |

Note: \* Adverse events are classified according to the MedDRA Version 21.1 by System Organ Class and Preferred Term.

Cohort Descriptions:

Mild: Subjects with mild renal impairment

Moderate: Subjects with moderate renal impairment Severe: Subjects with severe renal impairment Healthy: Healthy matched control subjects

TE = Treatment-emergent

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

CCI

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column. For each subject, please sort the AEs with same verbatim and preferred term by onset date/time. For any pair (e.g., AE\_S1, AE\_S2) of these AEs (for same subject, same verbatim and preferred term), if the onset date/time of AE\_S2 = resolved date/time of AE\_S1 and the grade of AE\_S2 < the grade level of AE\_S1, then mark the AE\_S2 with a flag like EVAUL\_FLG ="N". Then, for AE analysis (summary tables), please exclude the ones with EVAUL\_FLG ="N". Won't repeat this comment again.

Table 14.3.1.2 Treatment-emergent Adverse Event Frequency by Cohort - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

| | Cohort | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | N | <br>1ild | Mo | derate | | evere | | althy | 07 | verall |
| Number of TE Adverse Events | X | (100%) | | (100%) | | (100%) | | (100%) | | (100%) |
| Nervous system disorders | X | (XX%) | X | (XX%) | | (XX%) | | (XX%) | | (XX%) |
| Dizziness | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Headache | X | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Presyncope | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Respiratory, thoracic and mediastinal disorders | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Dry throat | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Oropharyngeal pain | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Sinus congestion | X | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Sneezing | X | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| General disorders and administration site conditions | X | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Fatigue | X | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| Thirst | Χ | (XX%) | X | (XX%) | Χ | (XX%) | X | (XX%) | Χ | (XX%) |
| etc. | | | | | | | | | | |

Note: \* Adverse events are classified according to the MedDRA Version 21.1 by System Organ Class and Preferred Term.

DDMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

Statistical Analysis Plan, 23 May 2019


TE = Treatment-emergent

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>


Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by Cohort, Severity Grade, and Relationship to Study Drug - Number of Subjects Reporting Events (Safety Population)

| | | Number of<br>Subjects with | | Se | verit | y Grade | Relationship to Study Drug | | |
|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | Cohort | Adverse Events | 1 | 2 | 3 | 4 | 5 | Related | Not Related |
| Dizziness | XXXX | X | Х | Х | Χ | Χ | Х | X | X |
| Dry eye | XXXX | X | X | X | X | X | X | X | X |
| Dry mouth | XXXX | X | X | X | X | X | X | X | X |
| _ | XXXX | X | X | X | X | X | X | X | X |
| Dry throat | XXXX | X | X | X | X | X | X | X | X |
| Ear pain | XXXX | X | X | X | X | X | X | X | X |
| Fatigue | XXXX | X | Χ | Χ | Χ | Χ | Χ | X | X |
| Mild RI Subjects | | XX | X | Х | X | Х | X | X | X |
| Moderate RI Subjec | cts | XX | X | X | X | X | X | X | X |
| Severe RI Subjects | 3 | XX | X | X | X | X | X | X | X |
| Healthy Matched Su | ıbjects | XX | X | X | X | X | X | X | X |
| Overall | - | XX | Χ | Χ | Χ | Χ | Χ | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately lifethreatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity.

When a subject experienced the same TEAE at more than one level of severity, only the most severe one was counted.

When a subject experienced the same TEAE at more than one level of drug relationship, only the one related to study drug was counted.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

CCI DDMMYYYY HH:MM


Table 14.3.1.4 Treatment-Emergent Adverse Event Frequency by Cohort, Severity Grade, and Relationship to Study Drug - Number of Adverse Events (Safety Population)

| | | Number of | | Se | verit | y Grade | Э | Relationshi | p to Study Drug |
|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | Cohort | Adverse Events | 1 | 2 | 3 | 4 | 5 | Related | Not Related |
| Dizziness | XXXX | X | X | X | X | X | X | X | X |
| Dry eye | XXXX | X | X | X | X | X | X | X | X |
| Dry mouth | XXXX | X | X | X | X | X | X | X | X |
| - | XXXX | X | X | X | X | X | X | X | X |
| Dry throat | XXXX | X | X | X | X | X | X | X | X |
| Ear pain | XXXX | X | X | X | X | X | X | X | X |
| Fatigue | XXXX | X | Χ | Χ | Χ | Χ | Χ | X | X |
| Mild RI Subjects | | XX | X | X | X | X | X | X | X |
| Moderate RI Subjec | cts | XX | X | X | X | X | X | X | X |
| Severe RI Subjects | 3 | XX | X | X | X | X | X | X | X |
| Healthy Matched Su | ubjects | XX | X | X | X | X | X | X | X |
| Overall | - | XX | Χ | Χ | Χ | Χ | Χ | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

Table 14.3.2.1 Serious Adverse Events (Safety Population)

| | | | | | On | set/Resolut | ion | | | | | | Relationship |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject | | Adverse | PT*/ | | | | | Severity | | | Action for | Other To Study |
| Cohort | . Number | TE?^ | Event | SOC | Day | Date | Time | Freq* | Grade | Ser* | Outcome | Study Drug | Action Drug |
| XXXX | XXX-XXX | Yes | XXXXXXX | , | | DDMMMYYYY/ | | Inter. | X | NS | Resolved | XXXXXXXXX | XXXXXX XXXXXXXX |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent; PT = Preferred Term; SOC = System Organ Class, Onset day is relative to Day 1.

Freq\* represents Frequency: SE = Single Episode, Inter. = Intermittent, Cont. = Continuous

Ser\* represents Serious: NS = Not Serious

Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

CCI DDMMYYYY HH:MM

Programmer Note: if there are no serious adverse events reported, there will be just one table (Table 14.3.2.1) with the statement "There was no serious adverse event recorded during the study."

Statistical Analysis Plan, 23 May 2019


#### Tables 14.3.4.2-14.3.4.3 will have the following format.

Page 1 of X Table 14.3.4.1 Out-of-Range Values and Unscheduled Results - Serum Chemistry (Safety Population)

| Cohort | Site-<br>Subject<br>Number | Age\$/<br>Sex | Visit | Time Point | Date | Parameter1<br>(Unit) | Parameter2<br>(Unit) | Parameter3<br>(Unit) | Parameter4<br>(Unit) | Parameter5<br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX-XXX | XX/M | XXXXX | | DDMMYYYY | XX HN | XX | XX | XX | XX HN |
| | | | XXXXX | XXXXXXX | DDMMYYYYY | XX | XX | XX | XX | XX |
| | | | XXXXX | XXXXXXX | DDMMYYYYY | XX | XX | XX | XX HN | XX |
| | | | | | DDMMYYYYY | XX | XX | XX | XX | XX |
| | | | | | DDMMYYYY | XX LY- | XX LN | XX | XX LY- | XX |

Programmer Notes: Clinical laboratory results will be presented in SI units. Please include flags as appropriate next to each value if present in the database and add a footer with the flag definition. The ranges will not be presented in the header given that there is more than one site involved in the study and the following footnote will be added: 'Refer to appendix 16.1.10.1 for site specific reference ranges.'. Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination records chronologically with other scheduled assessments. Arrange alphabetically by lab test name.

> Clinically significant lab values generally will be captured as AEs, some of which the PI may indicate in Appendix 16.2.8.1.6 lab comments (as per GPG.03.0028 sections 2.9 and 2.10). Derive an additional flag for PI flag -/+ based on comments (i.e. NCS/CS). Present this derived 4th column in all tables, and list only PI-determined out-of-range clinically significant lab values in Table 14.3.4.4.

Note: \$ Age is calculated from the date of dosing.

Abnormal flag: H = Above Reference Range, L = Below Reference Range

Computer Clinical significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Refer to appendix 16.1.10.1 for site specific reference ranges.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

Statistical Analysis Plan, 23 May 2019

DDMMMYYYY HH:MM


Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

| Cohort | Subject<br>Number | | | Time<br>Point | Date | Time | Department | Test | Result | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX-XXX | XX/X | XXXXX | XXXXX | DDMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX | X - X | mg/dL |
| | | | | | | | Serum Chemistry | | | | mg/dL |
| | | | XXXXX | XXXXX | DDMMYYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HY- | X - X | mg/dL |
| | | | XXXXX | XXXXX | DDMMYYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HN | X - X | mg/dL |

Programmer Notes: Clinical laboratory results will be presented in SI units. Please include flags as appropriate next to each value if present in the database and add a footer with the flag definition. All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table. If there were no CS values as deemed by PI (i.e., no "CS" or "Clinically Significant" in the PI comment field in the laboratory dataset), then this table will contain the following statement: "There were no laboratory values documented as clinically significant by the PI in the study."

Note: \$ Age is calculated from the date of dosing.

H = Above Reference Range, L = Below Reference Range

Computer: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

CC

#### Tables 14.3.5.1, 14.3.5.2, 14.3.5.4, 14.3.5.5, 14.3.5.7, and 14.3.5.8 will have the following format.


Table 14.3.5.1 Clinical Laboratory Summary - Serum Chemistry (Safety Population)

| | | | Cohort | | | |
|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Time<br>Point | Statistic | Mild | Modera | te Sever | e Healthy |
| Testname (unit) | Screening | n | X | X | Х | Х |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day -1 | n | X | Х | Х | Х |
| | _ | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day 2 | n | X | Х | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X . X |
| | | Maximum | XX | XX | XX | XX |

Programmer note: Similar for remaining laboratory tests. Sort alphabetically by lab test name. SI units will be used in the summarization of all clinical laboratory results. For the change from baseline tables, please remove the screening and Day -1 time points, keep the baseline definition footnote and change the 'Cohort' header to 'Change From Baseline'.

Note: Baseline is the last non-missing predose measurement prior to dosing (Day -1), including unscheduled assessments.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

DDMMYYYYY HH:MM

Statistical Analysis Plan, 23 May 2019


### Tables 14.3.5.3, 14.3.5.6, and 14.3.5.9 will have the following format:


Table 14.3.5.3 Clinical Laboratory Shift from Baseline - Serum Chemistry (Safety Population)

| | | Baseline L | | | Bas | eline | N | Baseline H | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory | Time | Р( | ostdos | e<br> | <br>F | ostdo | se | <br>Р | ostdo | se |
| Test (units) Cohort | Point | L | N | Н | L | N | Н | L | N | Н |
| Testname(unit) Mild | Day 2 | X | XX | X | Χ | XX | Х | Х | XX | Х |
| | Day 5 | X | XX | Χ | Χ | XX | Χ | Χ | XX | Х |
| | Day 8 | X | XX | Χ | Х | XX | Χ | X | XX | Χ |

Programmer note: Similar for remaining laboratory tests. Use N = Within Normal Range, O = Outside Normal Range for urinalysis shift table.

Note: N = Within Normal Range, L = Below Normal Range, H= Above Normal Range.

Baseline is the last non-missing predose measurement prior to dosing (Day -1), including unscheduled assessments.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

CC

### Tables 14.3.5.10 and 14.3.5.11 will have the following format:


Table 14.3.5.10 Vital Sign Summary (Safety Population)

| 7711 1 01 | m.' | | Cohort | | | |
|---|---|---|---|---|---|---|
| 9 | Time<br>Point | Statistic | Mild | Moderate Severe Health | | |
| Parameter1 (unit) | Screening | n | Х | Х | X | X |
| | | Mean | | | | |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day -1 | n | X | X | X | X |
| | | Mean | | | | |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X . X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day 1 Predose | n | X | X | X | X |
| | _ | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |

<Programmer note: Similar for remaining vital sign parameters and time points. For the change from baseline tables,
please remove the screening, Day -1, and Day 1 Predose time points, keep the baseline definition footnote and change
the 'Cohort' header to 'Change From Baseline'.</pre>

Note: Baseline is the last non-missing predose measurement prior to dosing (Day 1 Predose), including unscheduled assessments.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

DDMMYYYY HH:MM

Statistical Analysis Plan, 23 May 2019


### Tables 14.3.5.12 and 14.3.5.13 will have the following format:


Table 14.3.5.12 12-Lead Electrocardiogram Summary (Safety Population)

| Rec | W.' | Cohort | | | | |
|---|---|---|---|---|---|---|
| ECG<br>Parameter (unit) | Time<br>Point | Statistic | Mild | Modera | te Sever | e Healthy |
| Parameter1 (unit) | Screening | n | X | X | Х | Х |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day -1 | n | X | X | Х | X |
| | _ | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | Day 8 | n | X | X | Х | X |
| | - | Mean | X . X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |

Programmer note: Similar for remaining ECG parameters. For the change from baseline tables, please remove the Screening and Day -1 time points, keep the baseline definition footnote and change the 'Cohort' header to 'Change From Baseline'.

Note: Baseline is the last non-missing predose measurement prior to dosing (Day -1), including unscheduled assessments. All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

DDMMYYYY HH:MM

Statistical Analysis Plan, 23 May 2019


#### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final CSR. These listings will be generated off of the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New size font 9.

Note: The visit and time point variables will be presented as recorded in the datasets and can be added and removed as appropriate from the listings.

Appendix 16.1.7.2 Healthy Control Subjects Matched to Renal Function Groups

| Subject Number | Assigned Renal Function Group | Healthy MatchedSubject Number |
|---|---|---|
| XXX-XXX | XXXXXXXXX | XXX-XXX |
| XXX-XXX | XXXXXXXXX | XXX-XXX |
| XXX-XXX | XXXXXXXXX | XXX-XXX |
| XXX-XXX | XXXXXXXXXX | XXX-XXX |
| XXX-XXX | XXXXXXXXX | XXX-XXX |
| XXX-XXX | XXXXXXXXX | XXX-XXX |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Site | Laboratory Group | Test Name | Sex | Age<br>Category | Conventional<br>Normal Range | Conventional<br>Unit | SI<br>Normal Range | SI<br>Units |
|---|---|---|---|---|---|---|---|---|
| XXX | Serum Chemistry | Test Name Test Name Test Name Test Name Test Name Test Name Test Name | XXXXXX<br>XXXXXX<br>XXXXXX<br>XXXXXX<br>XXXXXX | XX<br>XX<br>XX<br>XX<br>XX<br>XX | XX - XX<br>XX - XX<br>XX - XX<br>XX - XX<br>XX - XX<br>XX - XX | units units units units units units units | XX - XX<br>XX - XX<br>XX - XX<br>XX - XX<br>XX - XX<br>XX - XX | units units units units units units units |
| | Hematology | Test Name Test Name Test Name Test Name Test Name | XXXXXX<br>XXXXXX<br>XXXXXX<br>XXXXXX | XX<br>XX<br>XX<br>XX<br>XX | XX - XX<br>XX - XX<br>XX - XX<br>XX - XX | units<br>units<br>units<br>units<br>units | XX - XX<br>XX - XX<br>XX - XX<br>XX - XX | units<br>units<br>units<br>units<br>units |

Programmer note: Sort alphabetically by lab test name within each lab group.

<similar for remaining Laboratory Groups and Test Names>

Appendix 16.2.1 Subject Discontinuation (Safety Population)

| Cohort | Site/<br>Subject<br>Number | Date of Study Completion<br>End of Study or Date of<br>Discontinuation | | Primary<br>Discontinuation Reason | Specify |
|---|---|---|---|---|---|
| XXXXXX | XXX-XXX | DDMMYYYY | YES | | |
| | XXX-XXX | DDMMYYYYY | YES | | |
| | XXX-XXX | DD <b>MM</b> YYYY | YES | | |
| | XXX-XXX | DDMMYYYYY | YES | | |
| | XXX-XXX | DDMMYYYYY | NO | Adverse Event | XXXXXXXXXX |
| | XXX-XXX | DDMMYYYY | YES | | |
| | XXX-XXX | DDMMYYYY | YES | | |
| | XXX-XXX | DDMMYYYYY | YES | | |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYYY HH:MM


#### Appendix 16.2.4.1 Demographics (Safety Population)

| | Site/<br>Subject<br>Number | Date of<br>Birth | Age*<br>(yrs) | Reproductiv<br>Status | e<br>Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m^2) | Informed<br>Consent<br>Signed Date | Protocol<br>Version |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXX-XXX<br>XXX-XXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX<br>XX | AAAAAAA<br>AAAAAAA<br>AAAAAAA<br>AAAAAAA | AAAAAA<br>AAAAAA<br>AAAAAA<br>AAAAAA | AAAAAAA<br>AAAAAAA<br>AAAAAAA<br>AAAAAAA | AAAAAAAAA<br>AAAAAAAAAA<br>AAAAAAAAAA<br>AAAAAAA | XXX<br>XXX<br>XXX<br>XXX | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | AAAAAAAA<br>AAAAAAAA<br>AAAAAAAA<br>AAAAAAAA |

Programmer note: Please also include re-consent signed date and re-consent version.

Note: \* Age is calculated from the date of dosing.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023

### Celerion, Clinical Study Report No. CA25886

Appendix 16.2.4.2 Physical Examination (Safety Population)


| Cohort | Site/<br>Subject<br>Number | Visit | Time<br>Point | Date | Body<br>System | Answer or<br>Result | Comment |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXX-XXX | XXXXX | XXXXXX | DDMMYYYY | Was PE performed?<br>General<br>HEENT<br>< > | Yes<br>Normal<br>Normal<br>< > | |
| | | XXXXX | XXXXX | DDMMYYYY | Was PE performed?<br>HEENT<br>< > | Yes<br>Normal<br>< > | |

Programmer Note: The 'comment' column will present any data that is recorded in the 'Reason not done' or 'If Abnormal, Specify' fields of the CRF.

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>


#### Appendix 16.2.4.3 Medical and Surgical History (Safety Population)

| | Site/<br>Subject | Any | Date | | | | | |
|---|---|---|---|---|---|---|---|---|
| Cohort | _ | History? | Category | Body system | Start | End | Ongoing? | Condition or Events |
| XXXXX | XXX-XXX | XXX | Medical<br>Surgical | XXXXXXXXXX | DDMMYYYY<br>DDMMYYYY | | YES | XXXXXXX XXXXXXX XXXXXXXX |
| | XXX-XXX | XXX | Medical | XXXXXXXXXX | DDMMMYYY | Z DDMMYYYY | NO | |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYYY HH:MM


Appendix 16.2.4.4 Assessment of Renal Function (Safety Population)

| | Ci+o/ | eGFR #1 | | | eGF | R #2 | | | e clearance | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Site/<br>Subject<br>Number | Date | Time | Value<br>(unit) | Date | Time | Value<br>(Unit) | Mean eGFR<br>(unit) | Date | Result<br>(Unit) | _ |
| XXXXX | XXX-XXX<br>XXX-XXX<br>XXX-XXX | DDMMYYYY<br>DDMMYYYY | HH:MM<br>HH:MM | XXXXX<br>XXXXX<br>XXXXX | DDMMYYYY<br>DDMMYYYYY<br>DDMMYYYYY | HH:MM<br>HH:MM | XXXXX<br>XXXXX<br>XXXXX | XXXXXX<br>XXXXXX<br>XXXXXX | DDMMYYYYY<br>DDMMYYYYY<br>DDMMMYYYY | XXXXX<br>XXXXX<br>XXXXX | _ |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYY HH:MM


Appendix 16.2.5.1 Subject Eligibility (Safety Population)

| Cohort | Site/<br>Subject<br>Number | Did subject meet all eligibility criteria? | Specify |
|---|---|---|---|
| XXXXXX | XXX-XXX | YES | |
| | XXX-XXX | NO | <pre><this column="" data="" if="" is="" only="" present="" presented=""></this></pre> |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023

Celerion, Clinical Study Report No. CA25886


Appendix 16.2.5.2 Test Compound Administration Times (Safety Population)

| Site/<br>Subject<br>Cohort Number | | | Was Subject Fasted for at least 2 hours prior to dosing? | Was LOXO-292<br>Administered | , | | ed Time | Dosage<br>(Unit) | Route | Formulation | on Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX XXX-XXX | XXXXX | XXXXX | XXXXXX | XXXXXXX | XXXXXXX DI | OMMYYYY | XX:XX | XXXXXXX | XXXXX | XXXXXXX | <pre><this column="" data="" if="" is="" only="" present="" prints=""></this></pre> |

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYY HH:MM


Appendix 16.2.5.3 PK Blood Draw Times and Protein Binding (Safety Population)

| Site/<br>Subject<br>Cohort Number | | Time Point | | Predose<br>Plasma Protein<br>Binding Sample? | | | Comments |
|---|---|---|---|---|---|---|---|
| XXXX XXX-XX | X XXXXX | XXXXXXXX | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | XXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | X:XX<br>X:XX | |

Programmer note: If appropriate, please add the 'flag for programming' column if present to the database.

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>


Appendix 16.2.5.4 Urine Collection Times (Safety Population)

#### Urine Collection

| | Site/<br>Subject | | | Sample | Start | t<br> | Stop | | Volume | Weight | Unable<br>to | Subject<br>is | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Number | Day | Hour | Collected? | Date | Time | Date | Time | (mL) | (g) | Void? | Anuric? | Comments |
| XXXX | XXX-XXX | XX<br>XX | XXXX | XXXX<br>XXXX | DDMMYYYY<br>DDMMYYYYY | X:XX:XX<br>X:XX:XX | DDMMYYYY<br>DDMMYYYYY | X:XX:XX<br>X:XX:XX | XXX | XXX | XXXXX | XXXXX | XXXXXXXXXXX |

Programmer note: If appropriate, please add the 'flag for programming' column if present to the database.

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>


Appendix 16.2.5.5 Follow-Up Phone Call (Safety Population)

| | Site/<br>Subject | Was a Telephone Call | _ | | Any AE Since | Any new concomitant medication or change in concomitant medication |
|---|---|---|---|---|---|---|
| Cohort | | Performed? (Yes/No) | | If No, Reason* | Last Visit? | Since last visit ? |
| XXXX | XXX-XXX | YES | DDMMYYYY | XXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXX |

Note: \* Reason options: 3 call attempts with no subject return call; Phone Disconnected; Wrong Number All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYYY HH:MM


Appendix 16.2.5.6 Prior and Concomitant Medications (Safety Population)

| | Site/<br>Subject<br>Number | | | Medication<br>(WHO* Term) | Dosage | Route | Start<br>Frequency Day/Date/Time | | | (If Due | | nuing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXX-XXX<br>XXX-XXX | No<br>Yes | Yes | None<br>ACETAMINOPHE<br>(ACETAMINOPHE | _ | BY MOUTH | AS NEEDED XX/DDMMYYYY/ HH:MM | XX/DDMMYYYY/<br>HH:MM | XXXXX | NA | NA | YES |

Note: \* Concomitant medications are coded with WHO Dictionary Version 01Sep2018 B3.

Start and stop day is relative to Day 1.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

| | TITT NO. |
|-----------|----------|
| DDMMMYYYY | HH:MM |

<sup>^</sup> Med = Medication; UNK = Unknown; AE = Adverse Event; MH = Medical History; NA = Not Applicable Prior medication was medication taken prior to study drug administration.

#### Appendix 16.2.7.1 Adverse Events (I of II) (Safety Population)

| | Site/<br>Subject | | Adverse Event/ | Time from<br>Last Dose | | Onset | | | Resolved | Duration | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Number | TE?^ | Preferred Term* | (DD:HH:MM) | Day | Date | Time | Day | Date | Time | (DD:HH:MM) |
| XXX | XXX-XXX | | None | | | | | | | | |
| | XXX-XXX | Yes | XXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |
| | | No | XXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

<sup>^</sup> TE = Treatment-emergent, Onset and resolved day is relative to Day 1.

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023

### Celerion, Clinical Study Report No. CA25886


#### Appendix 16.2.7.2 Adverse Events (II of II) (Safety Population)

| | Site/<br>Subject Treat | | Treat- Adverse | | Onset | | | | | | Action for | Other<br>Action | Relationship to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | _ | ment | Event | Day | Date ' | Γime | Freq* | Severity | Ser | * Outcome | Study Drug | Taken | Study Drug |
| XXXX | XXX-XXX | | None | | | | | | | | | | |
| | XXX-XXX | Χ | XXXXXXX | XX | DDMMYYYY | XX:XX | Inter. | Grade 1 | NS | Recovered or<br>Resolved | Dose Not Chang | ged XXXXXXXX | Not Related |

Note: Ser\* represents Serious: NS = Not Serious

Freq\* represents Frequency: SE = Single Episode, Inter. = Intermittent, Cont. = Continuous

Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately

life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Onset and resolved day is relative to Day 1.

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>


#### Appendix 16.2.7.3 Adverse Event Comments (Safety Population)

| | Site/ | | | Onset | | | Resolve | d | |
|---|---|---|---|---|---|---|---|---|---|
| | Subject Adverse | | | | | | | | |
| Cohort | Number | Event | Day | Date | Time | Day | Date | Time | Comments |
| XXXXX | XXX-XXX | DRY LIPS | XX | DDMMYYYY | X:XX | XX | DDMMYYYYY | X:XX | XXXXXXXXXXX |

Note: Onset and resolved day is relative to Day 1.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>


Appendix 16.2.7.4 Adverse Event Preferred Term Classification (Safety Population)

| | Site/ | | | | | Onset | |
|---|---|---|---|---|---|---|---|
| Cohort | Subject<br>Number | Adverse<br>Event | Preferred Term* | System Organ Class* | Day | Date | Time |
| XXXX | XXX-XXX | XXXXXX XXXXX XXXX XXXXX | XXXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX | DDMMYYYY | X:XX |

Note: \* Adverse events are classified to MedDRA Version 21.1 by System Organ Class and Preferred Term.
Onset day is relative to Day 1.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CCI DDMMYYYYY HH;MM
### Appendices 16.2.8.1.1-16.2.8.1.5 will have the following format.


Appendix 16.2.8.1.1.1 Clinical Laboratory Report - Serum Chemistry (Conventional Units) (Safety Population)

| Site/ Subject Age\$, Cohort Number Sex | | oint Date | Parameter1<br>(Unit) | Parameter2<br>(Unit) | Parameter3<br>(Unit) | Parameter4<br>(Unit) | Parameter5<br>(Unit) |
|---|---|---|---|---|---|---|---|
| XXXXX XXX-XXX XX/M | XXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX DDMMMYYYY | XX HN<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX HN | XX HN<br>XX<br>XX |

Programmer Notes: Please also include the following columns in the listings as appropriate for each department: 'Was Sample Collected?', 'If no, reason', 'Was the subject fasting?', 'Any clinically significant results?'. These columns will be presented before the individual test results. Clinical laboratory results will be presented in SI and conventional units. Please include flags as appropriate next to each value if present in the database and add a footer with the flag definition. The ranges will not be presented in the header since there is more than one site involved in the study and the following footnote will be added: 'Refer to appendix 16.1.10.1 for site specific reference ranges.'. Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments. The reproductive status will also be included in the serum FSH listings.

> Clinically significant lab values generally will be captured as AEs, some of which the PI may indicate in Appendix 16.2.8.1.6 lab comments (as per GPG.03.0028 sections 2.9 and 2.10). Derive an additional flag for PI flag (+) based on positive CS/Clinically Significant comments. Present this derived 4th column in all tables, and list only PI-determined out-of-range clinically significant lab values in Table 14.3.4.4. Arrange alphabetically by lab test name.

Note: \$ Age is calculated from the date of dosing.

H = Above Reference Range, L = Below Reference Range

Computer Clinical Significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Refer to appendix 16.1.10.1 for site specific reference ranges.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

### Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMYYYYY HH:MM


Appendix 16.2.8.1.6 Clinical Laboratory Report - Comments (Safety Population)

| Cohort | Subject<br>Number | Visit | Time<br>Point | Date | Department | Test | SI<br>Result | SI<br>Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXX-XXX | XXX | XXXXXX | DDMMYYYY | Other Tests | Fibrinogen | XXX | mg/dL | Not significant in the context of this study. |

Programmer Note: Results will be presented in SI units.

Note: All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast. Cohort Descriptions: <description>

CC DDMMYYYYY HH:MM

### Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886


Appendix 16.2.8.1.7 Clinical Laboratory Serology Samples (Safety Population)

| Site/<br>Subject<br>Cohort Number | Age\$/<br>Sex | Visit | Date | Was the Sample<br>Collected? |
|---|---|---|---|---|
| XXXXX XXX-XXX | XX/M | XXXXXX<br>XXXXXX<br>XXXXXX | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | XX<br>XX<br>XX |

Note: \$ Age is calculated from the date of dosing.

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

DDMMYYYY HH:MM

### Loxo Oncology, Inc. LOXO-292, LOXO-RET-18023 Celerion, Clinical Study Report No. CA25886


#### Appendix 16.2.8.2 Vital Signs (Safety Population)

| | | | | | | | | Blood Pressure (mmHg) | | Respir- | <ul> <li>Temper-</li> </ul> | - | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject | | Time | | | | Supine for | | Pulse | ation | ature | Weight | |
| Cohort | Number | Visit | Point | Date | Time | Position | at least 5 minutes? | Systolic/Diastolic | (bpm) | (rpm) | (°C) | (kg) | Comments |
| XXX | XXX-XXX | XXXXX | XXXXXX | DDMMYYYY | X:XX | | | | | | | XXX.X | |
| | | XXXXX | XXXXXX | DDMMYYYY | X:XX | SIT | XXXX | XXX/ XX | XX | XX | XX.X | | |
| | | XXXXX | XXXXXX | DDMMYYYYY | XX:XX | | | | | | | XXX.X | |
| | | XXXXX | XXXXXX | DDMMYYYY | XX:XX | SIT | XXXX | XXX/ XX | XX | XX | | | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Please also include 'Not Done' if populated by 'Yes' in the database. If appropriate, please add the 'flag for programming' column if present to the database.

Note: SIT = Sitting

All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.

Cohort Descriptions: <description>

CCI DDMMYYYY HH:MM


#### Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Cohort | Subject<br>Number | Visit | Time<br>Point | Date | Time | Was Subject<br>supine for at<br>least 10 minutes? | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | RR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF*<br>(msec) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXX-XXX | XXXXX<br>XXXXX<br>XXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | X:XX<br>X:XX<br>X:XX | XXX<br>XXX<br>XXX<br>XXX | Normal<br>ANCS<br>Normal<br>Normal | XX<br>XX<br>XX<br>XX | XXX.X<br>XXX.X<br>XXX.X | XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | XXX.X<br>XXX.X<br>XXX.X | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X # | |
| | | | XXXXXXX | DDMMYYYYY | X:XX | XXX | Normal | XX | XXX.X | XX.X | XX.X | XXX.X | XXX.X @ | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments. Please also include 'Not Done' if populated by 'Yes' in the database. If appropriate, please add the 'flag for programming' column if present to the database.

Note: ANCS = Abnormal, Not Clinically Significant
QTcF\* = QT corrected for heart rate using Fridericia's correction.
# = QTcF > 450, @ = QTcF change from baseline greater than 30 msec
All subjects received a single oral dose of 160 mg LOXO-292 following a 2-hour fast.
Cohort Descriptions: <description>

DDMMYYYY HH:MM

### **16.1.9.2** Statistical Outputs

# Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t for Table 14.2.1.10 (Paired t-test)

The TTEST Procedure

| | | Diff | erence: | Mild | - Healt | hy | |
|---|---|---|---|---|---|---|---|
| N | Me | an St | d Dev | Std | Err | Minimum | Maximum |
| 8 | 0.03 | 96 0 | .3774 | 0.1 | 334 | -0.4846 | 0.5254 |
| N | <i>l</i> ean | 90% CL | Mean | S | td Dev | 90% | CL Std Dev |
| 0.0 | 396 | -0.2132 | 0.2924 | E E | 0.3774 | 0.2 | 662 0.6782 |
| | | D | F t V | Value | Pr > | t | |
| | | | 7 | 0.30 | 0.7 | 752 | |



#### Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf for Table 14.2.1.10 (Paired t-test)

The TTEST Procedure

| | | Diffe | erence: | Mild - | - Healt | hy | | |
|---|---|---|---|---|---|---|---|---|
| N | Mea | an Sto | l Dev | Std 1 | Err | Mini | mum | Maximum |
| 8 | 0.03 | 78 0. | 3766 | 0.1 | 331 | -0.4 | 833 | 0.5235 |
| N | <i>M</i> ean | 90% CL | Mean | S | td Dev | | 90% CL | Std Dev |
| 0.0 | 0378 | -0.2144 | 0.2900 | | 0.3766 | 0 | 0.2656 | 0.6768 |
| | | DF | t Va | alue | Pr > | t | | |
| | | 7 | ( | 0.28 | 0.7 | 847 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: Cmax for Table 14.2.1.10 (Paired t-test)

The TTEST Procedure

| Difference: | Mild - | - Healthy |
|-------------|--------|-----------|
|-------------|--------|-----------|

| N | | Mean | Std | Dev | Std | Err | Mini | mum | Maximum |
|---|---|---|---|---|---|---|---|---|---|
| 8 | 0 | 2328 | 0. | 5220 | 0. | 1846 | -0.4 | 1454 | 1.1183 |
| | Mean | 9 | 90% CL | Mean | | Std Dev | | 90% CL | Std Dev |
| 0. | 2328 | -0 | .1169 | 0.5824 | 1 | 0.5220 | | 0.3682 | 0.9381 |
| | | | DF | t v | /alue | Pr > | t | | |
| | | | 7 | | 1.26 | 0.2 | 477 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t for Table 14.2.1.11 (Paired t-test)

The TTEST Procedure

| Difference: | Moderate | _ | Healthy |
|-------------|----------|---|---------|
|-------------|----------|---|---------|

| N | | Mean | Std | Dev | Sto | d Err | Min | imum | Maximum |
|---|---|---|---|---|---|---|---|---|---|
| 8 | 0. | 5415 | 0. | 5311 | 0. | .1878 | -0. | 3158 | 1.2106 |
| | Mean | | 90% CL 1 | Mean | | Std Dev | | 90% CL | Std Dev |
| 0. | 5415 | 0 | .1858 | 0.897 | 72 | 0.5311 | | 0.3746 | 0.9544 |
| | | | DF | t | Value | Pr > | t | | |
| | | | 7 | | 2.88 | 0. | 0235 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf for Table 14.2.1.11 (Paired t-test)

The TTEST Procedure

| Difference: | Moderate | Yang. | Healthy |
|-------------|----------|-------|---------|
| DITTELEUCE: | Moderate | _ | nealuiv |

| N | Mea | n Std | Dev | Std Err | Mini | mum | Maximum |
|----|-------|--------|--------|---------|--------|--------|---------|
| 8 | 0.543 | 4 0. | 5311 | 0.1878 | -0.3 | 3113 | 1.2110 |
| | Mean | 90% CL | Mean | Std I | )ev | 90% CL | Std Dev |
| 0. | .5434 | 0.1877 | 0.8992 | 0.53 | 311 | 0.3747 | 0.9545 |
| | | DF | t Va | alue Pr | > t | | |
| | | 7 | 2 | 2.89 | 0.0232 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: Cmax for Table 14.2.1.11 (Paired t-test)

The TTEST Procedure

Difference: Moderate - Healthy

| N | Mean | Std | Dev | Std Err | Min | imum | Maximum |
|------|--------|----------|--------|---------|--------|--------|---------|
| 8 | 0.4204 | 1. | 0211 | 0.3610 | -0. | 6931 | 2.5017 |
| Me | ean | 90% CL 1 | Mean | Std I | )ev | 90% CL | Std Dev |
| 0.42 | 204 - | 0.2635 | 1.1043 | 1.02 | 211 | 0.7203 | 1.8350 |
| | | DF | t Val | lue Pi | c > t | | |
| | | 7 | 1 | .16 | 0.2824 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t for Table 14.2.1.12 (Paired t-test)

The TTEST Procedure

| | | Diffe | rence: | Severe - | - Healt | hy | |
|----|------|---------|--------|----------|---------|---------|---------|
| N | Me | ean Sto | d Dev | Std E | cr | Minimum | Maximum |
| 7 | 0.20 | 045 0 | .5711 | 0.215 | 58 | -0.3914 | 0.9839 |
| | Mean | 90% CL | Mean | Sto | d Dev | 90% CL | Std Dev |
| 0. | 2045 | -0.2150 | 0.6239 | 0. | 5711 | 0.3942 | 1.0938 |
| | | Di | e t v | alue | Pr > | tl | |
| | | | 6 | 0.95 | 0.38 | 801 | |



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf for Table 14.2.1.12 (Paired t-test)

The TTEST Procedure

| | | Differe | ence: S | evere - He | ealthy | |
|----|-------|----------|---------|------------|----------|------------|
| N | Mean | n Std | Dev | Std Err | Minimum | Maximum |
| 7 | 0.216 | 7 0.! | 5742 | 0.2170 | -0.3721 | 0.9847 |
| | Mean | 90% CL 1 | Mean | Std De | ev 90% ( | CL Std Dev |
| 0. | 2167 | -0.2050 | 0.6385 | 0.574 | 12 0.39 | 64 1.0999 |
| | | DF | t Va | lue Pr | > t | |
| | | 6 | 1 | .00 | .3566 | |



## Statistical Comparisons of Pharmacokinetic Parameter: Cmax for Table 14.2.1.12 (Paired t-test)

The TTEST Procedure

Difference: Severe - Healthy

| N | | Mean | Std | Dev | sto | l Err | Min | imm | Maximum |
|---|---|---|---|---|---|---|---|---|---|
| 7 | -0. | 1780 | 0. | 6735 | 0. | 2546 | -1. | 4332 | 0.6119 |
| | Mean | | 90% CL | Mean | | Std Dev | | 90% CL | Std Dev |
| -0. | 1780 | -0 | .6727 | 0.3167 | | 0.6735 | | 0.4649 | 1.2901 |
| | | | DF | t V | alue | Pr > | t | | |
| | | | 6 | 4 | 0.70 | 0.5 | 105 | | |



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t,u for Table 14.2.3.14 (Paired t-test)

The TTEST Procedure

| | | | Diffe | rence: | Mild | - Healt | hy | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 1 | Mean | Std | Dev | Std | Err | Min | imum | Maxir | num |
| 8 | 3 0 | .0662 | 0. | 3302 | 0. | 1167 | -0. | 2769 | 0.64 | 132 |
| | Mean | 9 | 90% CL | Mean | | Std Dev | | 90% CL | Std De | ēν |
| | 0.0662 | -0. | 1550 | 0.2874 | | 0.3302 | | 0.2329 | 0.59 | 935 |
| | | | DF | t V | alue | Pr > | t | | | |

0.57

0.5886



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf,u for Table 14.2.3.14 (Paired t-test)

The TTEST Procedure

| | | Diffe | erence: | Mild - Healt | thy | |
|-----|--------|---------|---------|--------------|---------|---------|
| N | Mea | n Sto | l Dev | Std Err | Minimum | Maximum |
| 8 | 0.064 | 13 0. | 3298 | 0.1166 | -0.2794 | 0.6393 |
| 1 | Mean ( | 90% CL | Mean | Std Dev | 90% CL | Std Dev |
| 0.0 | 0643 | -0.1566 | 0.2853 | 0.3298 | 0.2327 | 0.5928 |
| | | DF | t Va | alue Pr > | [t] | |

0.55

0.5983



# Statistical Comparisons of Pharmacokinetic Parameter: Cmax,u for Table 14.2.3.14 (Paired t-test)

The TTEST Procedure

Difference: Mild - Healthy

| | | | | - | |
|---|--------|-------------|---------|---------|------------|
| N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 8 | 0.2593 | 0.5317 | 0.1880 | -0.4629 | 0.9349 |
| | Mean | 90% CL Mean | Std Dev | 90% | CL Std Dev |

DF t Value Pr > |t|
7 1.38 0.2102

0.5317 0.3751 0.9556

0.2593 -0.0969 0.6155



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t,u for Table 14.2.3.15 (Paired t-test)

The TTEST Procedure

| N Mean Std Dev Std Err Minimum M | aximum |
|------------------------------------|--------|
| 8 0.6333 0.5204 0.1840 -0.0706 | 1.3654 |
| Mean 90% CL Mean Std Dev 90% CL St | d Dev |
| 0.6333 0.2847 0.9819 0.5204 0.3671 | 0.9353 |
| DF t Value $Pr > t $ | |

3.44

0.0108



# Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf,u for Table 14.2.3.15 (Paired t-test)

The TTEST Procedure

| Difference: | Moderate | <ul> <li>Healthy</li> </ul> |
|-------------|----------|-----------------------------|
|-------------|----------|-----------------------------|

| N | Mear | n Std | Dev | Std E | rr | Minimum | n | Maximum |
|-----|--------|--------|--------|-------|-------|---------|------|---------|
| 8 | 0.6353 | 0. | 5202 | 0.18 | 39 | -0.0685 | 5 | 1.3653 |
| 1 | Mean | 90% CL | Mean | st | d Dev | 908 | cL S | Std Dev |
| 0.6 | 6353 | 0.2868 | 0.9837 | 0 | .5202 | 0.3 | 3669 | 0.9348 |
| | | DF | t V | alue | Pr > | t | | |
| | | 7 | | 3.45 | 0.0 | 106 | | |



# Statistical Comparisons of Pharmacokinetic Parameter: Cmax,u for Table 14.2.3.15 (Paired t-test)

The TTEST Procedure

| Difference: Modera | rate - Healthy |
|--------------------|----------------|
|--------------------|----------------|

| N | Mean | Std | Dev | Std Err | Minin | num | Maximum |
|---|---|---|---|---|---|---|---|
| 8 | 0.5122 | 1.0 | 0347 | 0.3658 | -0.56 | 527 | 2.4730 |
| Mea | n | 90% CL 1 | <b>M</b> ean | Std D | ev 9 | 90% CL | Std Dev |
| 0.512 | 2 -0 | .1809 | 1.2053 | 1.03 | 47 ( | .7299 | 1.8595 |
| | | DF | t Va | lue Pr | > t | | |
| | | 7 | 1 | .40 | 0.2042 | | |



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-t,u for Table 14.2.3.16 (Paired t-test)

The TTEST Procedure

| | | Differe | ence: S | Severe - | - Heal | thy | | |
|---|---|---|---|---|---|---|---|---|
| N | Mean | Std | Dev | Std E | rr | Mini | mum | Maximum |
| 7 | 0.4172 | 0. | 7358 | 0.278 | 31 | -0.2 | 507 | 1.5224 |
| 1 | Mean . | 90% CL 1 | <b>l</b> ean | Sto | d Dev | | 90% CL | Std Dev |
| 0.4 | 4172 - | 0.1233 | 0.9576 | 0. | 7358 | | 0.5079 | 1.4094 |
| | | DF | t Va | alue | Pr > | t | | |
| | | 6 | 1 | .50 | 0.1 | 843 | | |



## Statistical Comparisons of Pharmacokinetic Parameter: AUCO-inf,u for Table 14.2.3.16 (Paired t-test)

The TTEST Procedure

| | | | Differ | ence: | Sever | re - Heal | Lthy | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| N | | Mean | Std | Dev | Sto | l Err | Min | imum | Maximu | m |
| 7 | 0 | .4294 | 0. | 7403 | 0. | 2798 | -0. | 2414 | 1.562 | 2 |
| | Mean | | 90% CL | Mean | | Std Dev | | 90% CL | Std Dev | |
| 0 | .4294 | -0 | .1143 | 0.973 | 2 | 0.7403 | | 0.5111 | 1.418 | 1 |
| | | | DF | t | Value | Pr > | t | | | |
| | | | 6 | | 1.53 | 0.1 | 1758 | | | |



## Statistical Comparisons of Pharmacokinetic Parameter: Cmax,u for Table 14.2.3.16 (Paired t-test)

The TTEST Procedure

| | | Diffe | rence: | Severe | - Heal | thy | | |
|---|---|---|---|---|---|---|---|---|
| N | M | ean Sto | d Dev | Dev Std Er | | Minimum | | Maximum |
| 7 | 0.0 | 347 0 | .8208 | 0.3 | 102 | -1.2 | 926 | 0.9587 |
| 1 | <i>l</i> lean | 90% CL | Mean | S | td Dev | | 90% CL | Std Dev |
| 0.0 | 347 | -0.5682 | 0.6375 | 5 | 0.8208 | | 0.5666 | 1.5722 |
| | | Di | F t | <i>l</i> alue | Pr > | t | | |
| | | | 6 | 0.11 | 0.9 | 147 | | |



### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-t for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Residual
Residual
Residual
Residual
Residual

#### Class Level Information

| Class | Levels | Values |
|---------------|--------|------------|
| COHORT<br>SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 33 |

Cohort Descriptions:

A: Subjects with mild renal impairment B: Subjects with moderate renal impairment C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-t for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Number of Observations

| Number of Observations Read | 33 |
|---------------------------------|----|
| Number of Observations Used | 33 |
| Number of Observations Not Used | 0 |

#### Covariance Parameter Estimates

Cov Parm Estimate Residual 0.1767

#### Fit Statistics

| -2 Res Log Likelihood | 52.4 |
|--------------------------|------|
| AIC (Smaller is Better) | 54.4 |
| AICC (Smaller is Better) | 54.6 |
| BIC (Smaller is Better) | 55.7 |

Cohort Descriptions: A: Subjects with mild renal impairment B: Subjects with moderate renal impairment

rment

#### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-t for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.38 | 0.2697 |
| SEX | 1 | 26 | 4.76 | 0.0384 |
| AGE | 1 | 26 | 0.98 | 0.3312 |
| BMIBL | 1 | 26 | 0.39 | 0.5375 |

#### Estimates

| G0077E 15 | 600 UNE 1000 | Standard | | Eq. (SEREDONN) | | OKTEN DE | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| cohort A versus cohort D | 0.1993 | 0.2003 | 26 | 0.99 | 0.3289 | 0.1 | -0.1424 | 0.5410 |
| cohort B versus cohort D | 0.4060 | 0.2044 | 26 | 1.99 | 0.0577 | 0.1 | 0.05734 | 0.7546 |
| cohort C versus cohort D | 0.1103 | 0.2218 | 26 | 0.50 | 0.6233 | 0.1 | -0.2681 | 0.4886 |

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 10.1248 | 0.1512 | 26 | 66.98 | <.0001 | 0.1 | 9.8669 | 10.3826 |
| COHORT | В | 10.3315 | 0.1585 | 26 | 65.17 | <.0001 | 0.1 | 10.0611 | 10.6018 |
| COHORT | C | 10.0357 | 0.1704 | 26 | 58.91 | <.0001 | 0.1 | 9.7452 | 10.3263 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-t for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Least Squares Means

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Cohort | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| COHORT | D | 9.9255 | 0.1364 | 26 | 72.79 | <.0001 | 0.1 | 9.6929 | 10.1580 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



### Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Residual
Residual
Residual
Residual
Residual
Residual
Residual
Residual

#### Class Level Information

| Class | Levels | Values |
|---------------|--------|------------|
| COHORT<br>SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance : | Parameters | 1 |
|--------------|------------|----|
| Columns in 1 | X | 9 |
| Columns in | Z | 0 |
| Subjects | | 1 |
| Max Obs per | Subject | 33 |

### Cohort Descriptions:

A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Number of Observations

| Number of Observations Read | 33 |
|---------------------------------|----|
| Number of Observations Used | 33 |
| Number of Observations Not Used | 0 |

#### Covariance Parameter Estimates

Cov Parm Estimate Residual 0.1779

#### Fit Statistics

| -2 Res Log Likelihood | 52.6 |
|--------------------------|------|
| AIC (Smaller is Better) | 54.6 |
| AICC (Smaller is Better) | 54.8 |
| BIC (Smaller is Better) | 55.9 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



#### Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.36 | 0.2755 |
| SEX | 1 | 26 | 4.70 | 0.0395 |
| AGE | 1 | 26 | 1.05 | 0.3155 |
| BMIBL | 1 | 26 | 0.33 | 0.5695 |

#### Estimates

| Label | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| cohort A versus cohort D | 0.1969 | 0.2010 | 26 | 0.98 | 0.3364 | 0.1 | -0.1460 | 0.5397 |
| cohort B versus cohort D | 0.4065 | 0.2051 | 26 | 1.98 | 0.0581 | 0.1 | 0.05668 | 0.7563 |
| cohort C versus cohort D | 0.1184 | 0.2226 | 26 | 0.53 | 0.5994 | 0.1 | -0.2613 | 0.4980 |

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 10.1284 | 0.1517 | 26 | 66.77 | <.0001 | 0.1 | 9.8697 | 10.3871 |
| COHORT | В | 10.3381 | 0.1591 | 26 | 64.99 | <.0001 | 0.1 | 10.0668 | 10.6094 |
| COHORT | C | 10.0499 | 0.1709 | 26 | 58.80 | <.0001 | 0.1 | 9.7584 | 10.3415 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | D | 9.9315 | 0.1368 | 26 | 72.58 | <.0001 | 0.1 | 9.6982 | 10.1649 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: Cmax for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Model Information

Data Set

Dependent Variable
Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Residual
Residual
Residual
Residual
Residual
Residual
Residual
Residual

#### Class Level Information

| Class | Levels | Values |
|---------------|--------|------------|
| COHORT<br>SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 33 |

### Cohort Descriptions:

A: Subjects with mild renal impairment B: Subjects with moderate renal impairment C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma LOXO-292 Pharmacokinetic Parameter: Cmax for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Number of Observations

| Number of Observations Read | 33 |
|-----------------------------|--------|
| Number of Observations Used | 33 |
| Number of Observations Not | Used 0 |

#### Covariance Parameter Estimates

Cov Parm Estimate Residual 0.4786

#### Fit Statistics

| -2 Res Log Likelihood | 78.3 |
|--------------------------|------|
| AIC (Smaller is Better) | 80.3 |
| AICC (Smaller is Better) | 80.5 |
| BIC (Smaller is Better) | 81.6 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



#### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: Cmax for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.42 | 0.2596 |
| SEX | 1 | 26 | 3.34 | 0.0793 |
| AGE | 1 | 26 | 0.19 | 0.6679 |
| BMIBL | 1 | 26 | 1.11 | 0.3026 |

#### Estimates

| Label | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| cohort A versus cohort D | 0.5248 | 0.3297 | 26 | 1.59 | 0.1236 | 0.1 | -0.03759 | 1.0871 |
| cohort B versus cohort D | 0.2591 | 0.3364 | 26 | 0.77 | 0.4481 | 0.1 | -0.3147 | 0.8329 |
| cohort C versus cohort D | -0.1592 | 0.3651 | 26 | -0.44 | 0.6664 | 0.1 | -0.7819 | 0.4635 |

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 7.7901 | 0.2488 | 26 | 31.31 | <.0001 | 0.1 | 7.3657 | 8.2144 |
| COHORT | В | 7.5244 | 0.2609 | 26 | 28.84 | <.0001 | 0.1 | 7.0795 | 7.9694 |
| COHORT | C | 7.1061 | 0.2804 | 26 | 25.35 | <.0001 | 0.1 | 6.6279 | 7.5843 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Total Plasma IOXO-292 Pharmacokinetic Parameter: Cmax for Tables 14.2.1.13 - 14.2.1.15

#### The Mixed Procedure

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | D | 7.2653 | 0.2244 | 26 | 32.37 | <.0001 | 0.1 | 6.8825 | 7.6481 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




# Statistical Comparisons of Unbound Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-t,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

#### Model Information

Data Set WORK.MIXEDLOXO292LAUCLST
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Degrees of Freedom Method Residual

#### Class Level Information

| Class | Levels | Values |
|------------|--------|------------|
| COHORT SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 33 |

## Cohort Descriptions:

A: Subjects with mild renal impairment B: Subjects with moderate renal impairment C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-t,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

## Number of Observations

| Number of Observations Read | 33 |
|---------------------------------|----|
| Number of Observations Used | 33 |
| Number of Observations Not Used | 0 |

#### Covariance Parameter Estimates

Cov Parm **Estimate** Residual 0.2142

## Fit Statistics

| -2 Res Log Likelihood | 57.4 |
|--------------------------|------|
| AIC (Smaller is Better) | 59.4 |
| AICC (Smaller is Better) | 59.6 |
| BIC (Smaller is Better) | 60.7 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-t,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.40 | 0.2641 |
| SEX | 1 | 26 | 3.42 | 0.0757 |
| AGE | 1 | 26 | 2.77 | 0.1080 |
| BMIBL | 1 | 26 | 0.03 | 0.8656 |

## Estimates

| Label | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| cohort A versus cohort D | 0.2337 | 0.2206 | 26 | 1.06 | 0.2991 | 0.1 | -0.1425 | 0.6099 |
| cohort B versus cohort D | 0.4555 | 0.2251 | 26 | 2.02 | 0.0534 | 0.1 | 0.07161 | 0.8393 |
| cohort C versus cohort D | 0.2739 | 0.2442 | 26 | 1.12 | 0.2724 | 0.1 | -0.1427 | 0.6904 |

## Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 6.5687 | 0.1664 | 26 | 39.47 | <.0001 | 0.1 | 6.2849 | 6.8526 |
| COHORT | В | 6.7905 | 0.1745 | 26 | 38.91 | <.0001 | 0.1 | 6.4928 | 7.0882 |
| COHORT | C | 6.6089 | 0.1876 | 26 | 35.24 | <.0001 | 0.1 | 6.2890 | 6.9288 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-t,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | D | 6.3350 | 0.1501 | 26 | 42.20 | <.0001 | 0.1 | 6.0790 | 6.5911 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




# Statistical Comparisons of Unbound Plasma IOXO-292 Pharmacokinetic Parameter: AUCO-inf,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Residual
Residual
Residual
Residual
Residual
Residual
Residual
Residual

#### Class Level Information

| Class | Levels | Values |
|---------------|--------|------------|
| COHORT<br>SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 33 |

## Cohort Descriptions:

A: Subjects with mild renal impairment B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

## Number of Observations

| Number of Observations Read | 33 |
|-----------------------------|--------|
| Number of Observations Used | 33 |
| Number of Observations Not | Used 0 |

#### Covariance Parameter Estimates

Cov Parm **Estimate** Residual 0.2155

## Fit Statistics

| -2 Res Log Likelihood | 57.6 |
|--------------------------|------|
| AIC (Smaller is Better) | 59.6 |
| AICC (Smaller is Better) | 59.7 |
| BIC (Smaller is Better) | 60.8 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.40 | 0.2640 |
| SEX | 1 | 26 | 3.38 | 0.0775 |
| AGE | 1 | 26 | 2.87 | 0.1025 |
| BMIBL | 1 | 26 | 0.05 | 0.8331 |

## Estimates

| Label | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| cohort A versus cohort D | 0.2312 | 0.2213 | 26 | 1.05 | 0.3056 | 0.1 | -0.1461 | 0.6086 |
| cohort B versus cohort D | 0.4560 | 0.2258 | 26 | 2.02 | 0.0538 | 0.1 | 0.07092 | 0.8410 |
| cohort C versus cohort D | 0.2820 | 0.2450 | 26 | 1.15 | 0.2603 | 0.1 | -0.1359 | 0.6998 |

#### Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 6.5724 | 0.1670 | 26 | 39.37 | <.0001 | 0.1 | 6.2876 | 6.8571 |
| COHORT | В | 6.7971 | 0.1751 | 26 | 38.82 | <.0001 | 0.1 | 6.4985 | 7.0957 |
| COHORT | C | 6.6231 | 0.1881 | 26 | 35.20 | <.0001 | 0.1 | 6.3022 | 6.9440 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: AUCO-inf,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | D | 6.3411 | 0.1506 | 26 | 42.10 | <.0001 | 0.1 | 6.0843 | 6.5980 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




# Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: Cmax,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

#### Model Information

Data Set

Dependent Variable
Covariance Structure
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Residual
Residual
Residual
Residual
Residual
Residual
Residual
Residual

#### Class Level Information

| Class | Levels | Values |
|---------------|--------|------------|
| COHORT<br>SEX | 4 2 | ABCD<br>FM |

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 33 |

## Cohort Descriptions:

A: Subjects with mild renal impairment B: Subjects with moderate renal impairment C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: Cmax,u for Tables 14.2.3.17 - 14.2.3.19

#### The Mixed Procedure

## Number of Observations

| Number of Observations Read | 33 |
|---------------------------------|----|
| Number of Observations Used | 33 |
| Number of Observations Not Used | 0 |

#### Covariance Parameter Estimates

Cov Parm **Estimate** Residual 0.5746

## Fit Statistics

| -2 Res Log Likelihood | 83.1 |
|--------------------------|------|
| AIC (Smaller is Better) | 85.1 |
| AICC (Smaller is Better) | 85.2 |
| BIC (Smaller is Better) | 86.3 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment



#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: Cmax,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| COHORT | 3 | 26 | 1.03 | 0.3974 |
| SEX | 1 | 26 | 2.52 | 0.1247 |
| AGE | 1 | 26 | 0.75 | 0.3959 |
| BMIBL | 1 | 26 | 0.26 | 0.6150 |

## Estimates

| T-11 | 77 - 1 - 2 1 | Standard | DE | L **- 1 | De la IIII | 77-1- | ¥ | ** |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| cohort A versus cohort D | 0.5591 | 0.3612 | 26 | 1.55 | 0.1338 | 0.1 | -0.05701 | 1.1753 |
| cohort B versus cohort D | 0.3086 | 0.3686 | 26 | 0.84 | 0.4101 | 0.1 | -0.3201 | 0.9373 |
| cohort C versus cohort D | 0.004353 | 0.4000 | 26 | 0.01 | 0.9914 | 0.1 | -0.6779 | 0.6866 |

## Least Squares Means

| Effect | Cohort | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| COHORT | A | 4.2340 | 0.2726 | 26 | 15.53 | <.0001 | 0.1 | 3.7691 | 4.6990 |
| COHORT | В | 3.9835 | 0.2859 | 26 | 13.94 | <.0001 | 0.1 | 3.4959 | 4.4711 |
| COHORT | C | 3.6792 | 0.3072 | 26 | 11.98 | <.0001 | 0.1 | 3.1553 | 4.2032 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment




#### Statistical Comparisons of Unbound Plasma LOXO-292 Pharmacokinetic Parameter: Cmax,u for Tables 14.2.3.17 - 14.2.3.19

## The Mixed Procedure

## Least Squares Means

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Cohort | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| COHORT | D | 3.6749 | 0.2459 | 26 | 14.94 | <.0001 | 0.1 | 3.2555 | 4.0943 |

Cohort Descriptions:
A: Subjects with mild renal impairment
B: Subjects with moderate renal impairment

C: Subjects with severe renal impairment

